

Title: Nesina Tablets Special Drug Use Surveillance: Mild Type 2 Diabetes Mellitus

NCT Number: NCT01964963

Statistical analysis plan Approve Date: 04-Feb-2019

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

# Statistical Analysis Plan

# Nesina Tablets Special Drug Use Surveillance: Mild Type 2 Diabetes Mellitus

(Final Analysis)

Takeda Pharmaceutical Company Limited.
PPD

PPD

Version 3.0, Created on February 4, 2019

## Table of Contents

| 1.0 | Definition of Terms and Handling of Laboratory/Measured Data | 1 |
|---|---|---|
| 1.1 | Definitions | 1 |
| 1.2 | Important Identified Risks, Potential Risks, and Missing Information | .10 |
| 1.3 | Display digit | .11 |
| 1.4 | Level of Significance and Confidence Coefficient | .12 |
| 1.5 | Handling of Laboratory/Measured Data | .12 |
| 1.6 | Display Data Digit | .12 |
| 2.0 | Disposition of Patients (Patient Diagram) | .14 |
| 3.0 | Patient Demographics | .15 |
| 4.0 | Details of Treatment | .18 |
| 4.1 | Initial Dose of Nesina and Mean Daily Dose of Nesina, by Severity of Renal Impairment | .19 |
| 5.0 | Safety Tabulation and Analysis | .21 |
| 5.1 | Occurrence of adverse events and adverse drug reactions / infections | .21 |
| 5.1 | 1.1 Occurrence of adverse events | .21 |
| 5.1 | 1.2 Occurrence of adverse drug reactions / infections | .21 |
| 5.1 | 1.3 Important Identified Risks, Important Potential Risks, and Important Missing Information | .22 |
| 5.2 | Occurrence of Adverse Events and Adverse Drug Reactions / Infections in the Not Safety Analy | sis |
| Set | 23 | |
| 5.2 | 2.1 Occurrence of Adverse Events | .23 |
| 5.2 | 2.2 Occurrence of adverse drug reactions / infections | .24 |
| 5.3 | Occurrence of Adverse Drug Reactions / Infections by Severity, Onset Period, and Outcome | .25 |
| 5.3 | Occurrence of Adverse Drug Reactions / Infections by Severity, Onset Period, and Outcome | 25 |
| 5.4 | Patient Demographics and Frequency of Adverse Drug Reactions / Infections by Treatment | .26 |
| 5.4 | Patients demographics and Frequency of Adverse Drug Reactions / Infections by Treatment | .26 |
| 5.5 | Occurrence of Adverse Drug Reactions / Infections by Age | .27 |
| 5.6 | Occurrence of Adverse Drug Reactions / Infections by Sex | .28 |
| 5.7 | Occurrence of Adverse Drug Reactions / Infections by Liver Disorder | .28 |
| 5.8 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Renal Disorder | .28 |
| 5.9 | Occurrence of Adverse Drug Reactions / Infections by Severity of Renal Impairment | .29 |
| 5.10 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Heart Disease | .29 |
| 5.11 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Heart Failure | .29 |
| 5.12 | Occurrence of Adverse Drug Reactions / Infections by Severity of Heart Failure | .30 |
| 5.13 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Stroke-rela | ted |
| Disea | ase 30 | |
| 5.14 | Occurrence of Adverse Drug Reactions / Infections by Mean Daily Dose of Nesina | .30 |
| 5.15 | Occurrence of Adverse Drug Reactions / Infections by Mean Daily Dose of Nesina in Patients w | ith |
| Spec | ial Demographics (Patients with Moderate or Higher Renal Impairment) | .31 |
| 5.16 | Occurrence of Adverse Drug Reactions / Infections by Administration of Concomitant Medicat | ion |

| (Diabet | tic Drug) | 31 |
|---|---|---|
| 5.17 | Occurrence of Adverse Drug Reactions / Infections by Concomitant Medication (Diab | petic Drug) |
| | 31 | |
| 5.18 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concomitant | t Protease |
| Inhibite | ors | 32 |
| 5.19 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concomitant Rena | l Excretory |
| Drug | 32 | |
| 5.20 | Change in Laboratory/Measured Data | 32 |
| 5.20. | 1 Vital Signs | 32 |
| 5.20. | 2 Laboratory Values | 33 |
| 6.0 Ef | ficacy Tabulation and Analysis | 34 |
| 6.1 | Changes in HbA1c | 34 |
| 6.2 | Glycemic control achievement rate (HbA1c) | 34 |
| 6.3 | Changes in Fasting blood glucose level and Fasting insulin level | 34 |
| 6.4 | Changes in HbA1c, etc. by Factor Probably Affecting Efficacy | 35 |
| 6.5 | Changes in HbA1c, etc. in Patients with Special Demographics | 35 |

# 1.0 Definition of Terms and Handling of Laboratory/Measured Data

## 1.1 Definitions

| Term | Definition |
|---|---|
| Nesina | Nesina tablet(s) is abbreviated as Nesina in this statistical analysis plan. |
| SOC | System Organ Class of MedDRA/J |
| | MedDRA/J version 20.1 is used for this document. |
| HLGT | High level group term of MedDRA/J |
| PT | Preferred term of MedDRA/J |
| LLT | Lowest level term of MedDRA/J |
| Registered patients | Patients whose registration was approved |
| Survey sheet (electronic) | Patients whose survey sheets were sent via |
| collected patients | |
| Survey sheet (electronic) | Of the registered patients, patients whose survey sheets (electronic) were |
| uncollected patients | uncollected. |
| Safety Analysis Set | Of the survey sheet (electronic) collected patients, patients who were |
| | evaluated for safety analysis. |
| | For tabulation, the description of "total" means the Safety Analysis Set. |
| Not Safety Analysis Set | Of the survey sheet (electronic) collected patients, patients who were excluded |
| | from safety analysis |
| Efficacy Analysis Set | Of the Safety Analysis Set, patients who were evaluated for efficacy analysis |
| Not Efficacy Analysis Set | Of the Safety Analysis Set, patients who were excluded from the efficacy |
| | analysis |
| First date of Nesina | Of the start dates of the Nesina treatment period in patients, the earliest date is |
| treatment | defined as the first date of Nesina treatment. |
| Last date of Nesina | Of the last dates of the Nesina treatment period in patients, the latest date is |
| treatment | defined as the last date of Nesina treatment. If Nesina treatment is continued |
| | and the year, month, and date of the continued treatment period are specified, |
| | the year, month, and date of the continued treatment period are defined as the |
| | last date of Nesina treatment. If the data for the year, month, and date of the |
| | continued treatment period are missing, the following date is defined as the |
| | last date of Nesina treatment. |
| | (1) First date of Nesina treatment + 3 years (same month and date), if Nesina |
| | treatment is continued based on the survey sheet (electronic) after 36 |
| | months of treatment* |
| | (2) For other than the above, the first date of Nesina treatment + 1 year (same |
| | month and date), if Nesina treatment is continued based on the survey |
| | sheet (electronic) after 12 months of treatment** |

| Term | Definition |
|---|---|
| | For the continued treatment of Nesina, the following is considered as the "treatment to be continued:" • [End of Nesina tablet treatment] * If "No" for "Did you discontinue Nesina tablets by 12 to 36 months after the start of treatment?" ** If "No" for "Did you discontinue Nesina tablets by 12 months after |
| | the start of treatment?" |
| Adverse drug reactions, etc. | Abbreviation of "adverse drug reactions / infections" Of the adverse events, events for which causal relationship to Nesina was assessed as "Not related" by the Investigator. In this statistical analysis plan, "adverse drug reactions / infections" is used in the headings, while "adverse drug reactions, etc." is used in the sentences and tables. |
| Serious adverse events | Adverse events assessed as "serious" by the Investigator. Events described in the MedDRA coding list in the Takeda Medically Significant AE List will be handled as serious even if the Investigator assesses as "Not serious." |
| Serious adverse drug reactions | Abbreviation of "serious adverse drug reactions / infections" Of the "serious adverse events," the events for which causal relationship to Nesina was assessed as "Not related" by the Investigator |
| Number of patients with events | Number of patients with adverse events or adverse drug reactions, etc. |
| Number of events | Number of adverse events or adverse drug reactions, etc. |
| Percent of patients with events | [For safety analysis calculation in the Safety Analysis Set] The formula is: Number of patients with events / Number of Safety Analysis Set × 100. [For safety analysis calculation in the Not Safety Analysis Set] The formula is: Number of patients with events / Number of Not Safety |
| | Analysis Set × 100. |
| Percent of events | [For safety analysis calculation in the Safety Analysis Set] The formula is: Number of events / Number of the Safety Analysis Set × 100. [For safety calculation in the Not Safety Analysis Set] The formula is: Number of events / Number of Not Safety Analysis Set × 100. |
| Onset period | The formula is: Onset date of adverse events (or adverse drug reactions, etc.) – start date of Nesina treatment + 1. |

| Term | Definition |
|---|---|
| | For unknown onset date of adverse events (or adverse drug reactions, etc.), the |
| | onset period will be calculated as 1 day. However, if the start month and date |
| | of Nesina treatment are same as the onset month and date of adverse events |
| | (or adverse drug reactions, etc.), the onset period will be calculated as the start |
| | date of Nesina treatment. |
| Mild type 2 diabetes | Patients who have type 2 diabetes mellitus with HbA1c (NGSP value) of $\leq$ |
| mellitus | 7.4% at the start date of Nesina treatment |
| Patients with diabetic | Patients with any of the following complications: diabetic nephropathy, |
| complication | diabetic retinopathy, or diabetic neuropathy. |
| Patients with diabetic | Patients with complication of PT Code 10012660 (diabetic end stage renal |
| nephropathy | disease) or 10061835 (diabetic nephropathy). |
| Patients with diabetic | Patients with complication of PT Code 10012688 (diabetic retinal oedema) or |
| retinopathy | 10012689 (diabetic retinopathy). |
| Patients with diabetic | Patients with complication of PT Code 10012645 (diabetic autonomic |
| neuropathy | neuropathy), 10012676 (diabetic mononeuropathy), or 10012680 (diabetic |
| | neuropathy). |
| Patients with concurrent | Patients with concurrent disease of the Standardised MedDRA Query |
| hypertension | (hereinafter SMQ) Code 20000147 (hypertension (SMQ) narrow). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000026 (dyslipidaemia |
| dyslipidemia | (SMQ) narrow). |
| Patients with concurrent | Patients with concurrent disease of the PT code meeting the Takeda MedDRA |
| hyperuricemia | Query 20.1 (hereinafter, TMQ 20.1) (blood uric acid increased). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000005 (hepatic |
| liver disorder | disorders (narrow)). |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10019708 (hepatic steatosis). |
| hepatic steatosis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10019728 (hepatitis |
| alcoholic hepatitis | alcoholic). |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10008909 (chronic hepatitis). |
| chronic hepatitis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10019641 (hepatic cirrhosis). |
| hepatic cirrhosis | |
| Patients with concurrent | Patients with concurrent disease of the TMQ 20.1 (renal disease). |
| renal disorder | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10029164 (nephrotic |
| nephrotic syndrome | syndrome). |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10018364 |
| glomerulonephritis | (glomerulonephritis) or the PT Code 10018367 (glomerulonephritis chronic). |

| Term | Definition |
|---|---|
| Patients with concurrent | Patients with concurrent disease of the PT Code 10064848 (chronic kidney |
| chronic renal failure | disease) or the PT Code 10038435 (renal failure). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10007541 (cardiac |
| heart disease | disorders). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000004 (cardiac failure |
| cardiac failure | (SMQ) narrow). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000047 (myocardial |
| myocardial infarction | infarction (SMQ) narrow). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10007541 (cardiac |
| angina pectoris | disorders) and the PT Code 10036759 (prinzmetal angina), PT Code 10002383 |
| | (angina pectoris), PT Code 10058144 (postinfarction angina), PT Code |
| | 10002388 (angina unstable), or LLT Code 10065566 (microvascular angina). |
| Patients with concurrent | Patients with concurrent disease of cerebral infarction, cerebral haemorrhage, |
| stroke-related disease | subarachnoid haemorrhage, or transient ischaemic attack, described below. |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029205 (nervous system |
| disease cerebral infarction | disorders) and the PT Code 10006147 (brain stem infarction), PT Code |
| | 10008118 (cerebral infarction), PT Code 10008119 (cerebral infarction foetal), |
| | PT Code 10008034 (cerebellar infarction), PT Code 10019005 (haemorrhagic |
| | cerebral infarction), PT Code 10051078 (lacunar infarction), PT Code |
| | 10056237 (migrainous infarction), PT Code 10058571 (spinal cord infarction), |
| | PT Code 10060839 (embolic cerebral infarction), PT Code 10060840 |
| | (ischaemic cerebral infarction), PT Code 10064961 (thalamic infarction), PT |
| | Code 10067347 (thrombotic cerebral infarction), or PT Code 10069020 (basal |
| | ganglia infarction). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029205 (nervous system |
| cerebral hemorrhage | disorders) and the PT Code 10006145 (brain stem haemorrhage), PT Code |
| | 10008111 (cerebral haemorrhage), PT Code 10008112 (cerebral haemorrhage |
| | neonatal), PT Code 10008030 (cerebellar haemorrhage), PT Code 10018985 |
| | (haemorrhage intracranial), PT Code 10022840 (intraventricular |
| | haemorrhage), PT Code 10022841 (intraventricular haemorrhage neonatal), |
| | PT Code 10042365 (subdural haemorrhage neonatal), PT Code 10049236 |
| | (spinal epidural haemorrhage), PT Code 10048992 (spinal cord haemorrhage), |
| | PT Code 10050157 (cerebral haemorrhage foetal), PT Code 10052593 |
| | (meningorrhagia), PT Code 10058939 (thalamus haemorrhage), PT Code |
| | 10058940 (putamen haemorrhage), PT Code 10067057 (basal ganglia |
| | haemorrhage), PT Code 10067277 (cerebral microhaemorrhage), PT Code |
| | 10071205 (brain stem microhaemorrhage), PT Code 10071206 (cerebellar |
| | microhaemorrhage), PT Code 10072043 (central nervous system |

| Term | Definition |
|---|---|
| | haemorrhage), or PT Code 10073563 (Spinal subdural haemorrhage). |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10042316 (subarachnoid |
| subarachnoid hemorrhage | haemorrhage), PT Code 10042317 (subarachnoid haemorrhage neonatal), PT |
| | Code 10073564 (spinal subarachnoid haemorrhage), LLT Code 10072201 |
| | (Asymptomatic subarachnoid haemorrhage). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029205 (nervous system |
| transient ischemic attack | disorders) and the PT Code 10044390 (transient ischaemic attack). |
| Patients with concurrent | Patients with concurrent disease of bronchial asthma, pollinosis, allergic |
| allergic disease | rhinitis, or allergic dermatitis, described below. |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10038738 (respiratory, |
| bronchial asthma | thoracic and mediastinal disorders) and the PT Code 10003553 (asthma), PT |
| | Code 10075084 (aspirin-exacerbated respiratory disease), PT Code 10003557 |
| | (asthma exercise induced), PT Code 10003559 (asthma late onset), PT Code |
| | 10041961 (status asthmaticus), PT Code 10001890 (alveolitis allergic), PT |
| | Code 10049585 (infantile asthma), PT Code 10070836 (occupational asthma), |
| | or PT Code 10064823 (asthmatic crisis). |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10048908 (seasonal allergy). |
| pollinosis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10039085 (rhinitis allergic). |
| allergic rhinitis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10012434 (dermatitis |
| allergic dermatitis | allergic). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029104 (neoplasms |
| malignant tumor | benign, malignant and unspecified (incl cysts and polyps)). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000194 (malignant |
| malignant tumor (narrow | tumour (SMQ) narrow). |
| sense) | |
| Patients with other | Patients with concurrent disease other than the above (diabetic complication, |
| concurrent disease | hypertension, dyslipidaemia, hyperuricaemia, liver disease, renal disease, |
| | heart disease, stroke-related disease, allergic disease, malignant tumor, or |
| | malignant tumor (narrow sense)). |
| Severity of renal | Severity of renal impairment in the patient demographic section |
| impairment | |

| Term | Definition |
|---|---|
| Age | If the start month and date of Nesina treatment is earlier than the birth month |
| | and date, calculate using the following formula: Start year of Nesina treatment |
| | - birth year $-$ 1. If the birth month and date is earlier than or equal to the start |
| | month and date of Nesina treatment, calculate using the following formula: |
| | Start year of Nesina treatment – birth year. For unknown birth date, the birth |
| | date will be calculated as the 1st day of the birth month. |
| BMI | Calculate using the following formula: Weight (kg) / (0.0001 $\times$ Height (cm) $\times$ |
| | Height (cm)). Indicate to one decimal place rounded from two decimals. |
| Disease duration of type 2 | Calculate using the following formula: (start date of Nesina treatment - |
| diabetes mellitus (year) | diagnosis period of type 2 diabetes mellitus + 1) / 365.25. |
| | For unknown diagnosis month, calculate as January. |
| | Indicate to one decimal place rounded from two decimals. |
| Prior medication | Medications that patients were taking within 3 months before initiation of |
| | Nesina therapy. |
| Concomitant medication | Medications that patients were taking after the start date of Nesina treatment. |
| Start date of other diabetic | Calculate as the start date of survey sheet (electronic). |
| drug and concomitant | |
| medication (other than | |
| diabetic drug) | |
| End date of other diabetic | Calculate as the end date of survey sheet (electronic). |
| drug and concomitant | |
| medication (other than | |
| diabetic drug) | |
| Diabetic drugs | Drugs of the National Health Insurance (NHI) Drug List Code starting with |
| | 3969, 3961, 3962, 2492, 2499410, 2499411, 2499415, or 2499416. |
| α-glucosidase inhibitors | Drugs of the NHI Drug List Code starting with 3969003, 3969004, 3969009, |
| | or 3969102. |
| Thiazolidines | Drugs of the NHI Drug List Code starting with 3969005, 3969007, 3969100, |
| | 3969101, or 3969103. |
| Sulfonylureas | Drugs of the NHI Drug List Code starting with 3961 or 3969101. |
| Biguanides | Drugs of the NHI Drug List Code starting with 3962, 3969100, 3969104, or |
| | 3969105. |
| Rapid-acting insulin | Drugs of the NHI Drug List Code starting with 3969006, 3969008, 3969013, |
| secretagogues | or 3969102. |
| Insulin preparations | Drugs of the NHI Drug List Code starting with 2492. |
| DPP-4 inhibitors | Drugs of the NHI Drug List Code starting with 3969010, 3969011, 3969012, |
| | 3969014, 3969015, 3969016, 3969017, 3969024, 3969025, 3969103, |
| | 3969104, or 3969105. |
| ı | - |

| Term | Definition |
|---|---|
| GLP-1 receptor agonists | Drugs of the NHI Drug List Code starting with 2499410, 2499411, 2499415, |
| | or 2499416. |
| SGLT2 inhibitors | Drugs of the NHI Drug List Code starting with 3969018, 3969018, 3969019, |
| | 3969020, 3969021, 3969022, or 3969023. |
| Combination of diabetic | Drugs of the NHI Drug List Code starting with 3969100, 3969101, 3969102, |
| drugs | 3969103, 3969104, or 3969105. |
| Other diabetic drugs | Other diabetic drugs not classified into the above diabetic drug categories ( $\alpha$ - |
| | glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting |
| | insulin secretagogues, insulin preparations, DPP-4 inhibitors, GLP-1 receptor |
| | agonists, SGLT2 inhibitors, or combination of diabetic drugs). |
| Hypertension drugs | ARB Drugs of the NHI Drug List Code starting with the following 7 |
| | numbers: |
| | 2149039, 2149040, 2149041, 2149042, 2149044, 2149046, 2149048, |
| | 2149100, 2149110, 2149111, 2149112, 2149113, 2149114, 2149115, 2149116, |
| | 2149117, 2149118, 2149119, 2149120, 2149121, 2149122 |
| | Ca antagonists Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 2149019, 2149022, 2149027, 2149030, 2149034, 2149035, 2149037, |
| | 2149038, 2149043, 2149400, 2171006, 2171014, 2171019, 2171020, |
| | 2171021, 2171022, 2171405, 2190001, 2149114, 2149115, 2149116, |
| | 2149117, 2149118, 2149120, 2149121, 2149122, 2190101, 2190102, |
| | 2190103, 2190104 |
| | ACE inhibitors Drugs of the NHI Drug List Code starting with the following |
| | 4 numbers: |
| | 2144 |
| | Diuretics Drugs of the NHI Drug List Code starting with numbers 213 or the |
| | following 7 numbers: |
| | 2149003, 2149007, 2149012, 2149110, 2149111, 2149112, 2149113, |
| | 2149119, 2149122 |
| | α blockers Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 1234400, 214200210, 2149002, 2149015, 2149023, 2149026, 1152, 1149107, |
| | 1149114, 1149115, 2531001, 2149020 |
| | $\alpha\beta/\beta$ blockers $\;\;$ Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 2149032, 2149018, 2123014, 2149009, 2123013, 2123003, 2149008, |
| | 2149016, 2442001, 2123011, 2149036, 2123016, 2149700, 2149031, |
| | 2149010, 2123001, 2123F01, 2149029, 2123008, 2149014, 2149021, |

| Term | Definition |
|---|---|
| | 2149028, 2123015, 2123005, 2149025, 2123009, 2123403, 2149033, 2149011 |
| | Complication of hypertension drugs Drugs of the NHI Drug List Code |
| | starting with the following numbers: |
| | 2149110, 2149111, 2149112, 2149113, 2149114, 2149115, 2149116, 2149117, |
| | 2149118, 2149119, 2149120, 2149121, 2149122Other Drugs of the NHI Drug |
| | List Code starting with the following numbers: |
| | 2149047, 2142004, 2149001, 2149017, 2145 |
| Dyslipidaemia drugs | Statins Drugs of the NHI Drug List Code starting with the following numbers: |
| | 2189010, 2189011, 2189012, 2189013, 2189015, 2189016, 2189017, |
| | 2190101, 2190102, 2190103, 2190104 |
| | Fibrates Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 2183001, 2183002, 2183003, 2183004, 2183005, 2183006 |
| | EPA/DHA Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 2189019, 3399004 |
| | Other Drugs of the NHI Drug List Code starting with the following numbers: |
| | Dugs, other than the above, of the NHI Drug List Code starting with 218, |
| | 2900002, or 3133001. |
| Concomitant medication | Drugs other than the above (diabetic drugs, hypertension drugs, or |
| (other) | dyslipidaemia drugs). |
| Protease Inhibitor | Use the results of the drug name in the survey sheet (electronic) coded with |
| | the NHI Drug List (Appendix 1. List of Protease Inhibitors). |
| Renal excretory drugs | Use the results of the drug name in the survey sheet (electronic) coded with |
| | the NHI Drug List (Appendix 2. List of Renal Excretory Drugs). |
| Nesina treatment period | Actual treatment period from the start date to the end date of Nesina treatment. |
| (days) | However, the washout period is excluded from the treatment period. |
| | Calculate using the following formula: End of Nesina treatment – start date of |
| | Nesina treatment + 1 (grand total). |
| | (Consider the washout period.) |
| Mean daily dose of Nesina | Calculate using the following formula: Total of "daily dose of Nesina × Nesina |
| | treatment period at the relevant dose" / Nesina treatment period. For the |
| | calculation of Nesina treatment period, refer to the above. |
| | If the daily dose of Nesina is a number outside specification in the survey sheet |
| | (electronic) and is actual number, use the relevant number. |

| Term | Definition |
|---|---|
| HbA1c (NGSP value) | The NGSP value only will be used in this analysis. |
| | For the HbA1c (JDS value), calculate using the following formula: |
| | NGSP value (%) = $1.02 \times JDS$ value (%) + $0.25\%$ |
| | The HbA1c (international standard value) will be handled as the NGSP value. |
| Change in HbA1c | For HbA1c converted to the NGSP value, calculate using the following |
| | formula: Laboratory value - Laboratory value at the start of Nesina |
| | treatment. |
| Glycemic control | Divide the following two categories for the Glycemic control achievement |
| achievement rate | rate: |
| | HbA1c (NGSP converted value) [Unit %] |
| | NGSP (%): < 6.0, ≥6.0 / < 7.0,≥ 7.0 |
| non-HDL cholesterol | Calculate using the following formula: "Total cholesterol" - "HDL |
| | cholesterol." |
| Summary statistics | Number of patients, mean, standard deviation, minimum, first quartile, |
| | median, third quartile, and maximum. |

## 1.2 Important Identified Risks, Potential Risks, and Missing Information

| Term | Definition |
|---|---|
| Important identified risk | |
| Hypoglycemia | Adverse events of the following PT Codes (term) are defined as hypoglycemia. |
| | 10020994(Hypoglycaemia neonatal) |
| | 10040576(Shock hypoglycaemic) |
| | 10021000(Hypoglycaemic coma) |
| | 10020993(Hypoglycaemia) |
| | 10065981(Hypoglycaemic unconsciousness) |
| | 10021002(Hypoglycaemic encephalopathy) |
| | 10048803(Hypoglycaemic seizure) |
| | 10020997(Hypoglycaemia unawareness) |
| | 10077216(Hyperinsulinaemic hypoglycaemia) |
| | 10059035(Postprandial hypoglycaemia) |
| Acute pancreatitis | Adverse events of the SMQ Code 20000022 (acute pancreatitis (SMQ) narrow |
| | scope are defined as acute pancreatitis. |
| Hepatic impairment / | Adverse events of the SMQ Code 20000005 (hepatic disorders (SMQ) broad) |
| jaundice | are defined as hepatic impairment / jaundice. |
| Skin disorder including | Adverse events of the SMQ Code 20000020 (severe skin adverse reactions |
| oculomucocutaneous | (SMQ) narrow) are defined as skin disorder including oculomucocutaneous |
| syndrome (Stevens- | syndrome (Stevens-Johnson syndrome) / erythema multiforme. |
| Johnson syndrome) / | |
| erythema multiforme | |
| Rhabdomyolysis | Adverse events of the SMQ Code 20000002 (rhabdomyolysis/myopathy |
| | (SMQ) narrow) are defined as rhabdomyolysis. |
| Intestinal obstruction | Adverse events of the SMQ Code 20000105 (gastrointestinal obstruction |
| | (SMQ) narrow) or the HLGT Code 10018008 (gastrointestinal stenosis and |
| | obstruction) or HLT Code 10052736 (non-mechanical ileus) are defined as |
| | intestinal obstruction. |
| Interstitial pneumonia | Adverse events of the SMQ Code 20000042 (interstitial lung disease (SMQ) |
| | narrow) are defined as interstitial pneumonia. |
| Angioedema | Adverse events of the SMQ Code 20000024 (angioedema (SMQ) narrow) are |
| | defined as angioedema. |
| Important potential risk | |
| Infection | Adverse events of SOC Code 10021881(infections and infestations) are |
| | defined as infection. |
| Malignant tumor | Adverse events of the SOC Code 10029104 (neoplasms benign, malignant |
| | and unspecified (incl cysts and polyps)) are defined as malignant tumor. |
| Malignant tumor (narrow | Adverse events of the SMQ Code 20000194 (malignant tumors (SMQ) |

| Term | Definition |
|---|---|
| sense) | narrow) are defined as malignant tumor (narrow sense). |
| Pemphigoid | Adverse events of the PT Code 10067776 (ocular pemphigoid) or 10034277 |
| | (pemphigoid) are defined as pemphigoid. |

| Term | Definition |
|---|---|
| Important missing | |
| information | |
| Cardiovascular system risk | Adverse events of the SMQ Code 20000047 (myocardial infarction (SMQ) |
| | broad) or SMQ Code 20000061 (central nervous system haemorrhages and |
| | cerebrovascular conditions (SMQ) broad) are defined as cardiovascular |
| | system risk. |
| | "Central nervous system haemorrhage and cerebrovascular conditions (SMQ) |
| | broad" includes the following SMQ classes. |
| | > 20000166(Conditions associated with central nervous system |
| | haemorrhages and cerebrovascular accidents (SMQ) broad) |
| | > 20000064(Cerebrovascular disorder haemorrhagic (SMQ) |
| | broad) |
| | > 20000063(Cerebrovascular disease ischaemic (SMQ) broad) |

# 1.3 Display digit

| Term | Definition |
|---|---|
| Percentage (%) | Percent of patients with adverse events or adverse drug reactions, etc. or percent |
| | of adverse events or adverse drug reactions, etc.: |
| | Indicate to two decimal places rounded from three decimals. |
| | Other than the above: |
| | Indicate to one decimal place rounded from two decimals. |
| Summary statistics | Mean, median, first quartile, and third quartile: |
| | Indicate one lower digit rounded from two lower digits than the digit of the |
| | to-be evaluated data. |
| | Standard deviation: |
| | Indicate two lower digits rounded from three lower digits of the to-be |
| | evaluated data. |
| | Minimum and maximum |
| | Indicate the same digit number as that of the to-be evaluated data (refer to |
| | <u>Section 1.6</u> ). |
| p-value | Indicate to three decimal places rounded down from four decimals. |

| Term | Definition |
|---|---|
| | If the data is rounded down from four decimal places and less than 0.001, display |
| | as $p < 0.001$ . |

## 1.4 Level of Significance and Confidence Coefficient

Two-sided 5%, two-sided 95%.

## 1.5 Handling of Laboratory/Measured Data

- VISIT as described in the survey sheet will be used for data other than 12 months and 36 months after
   Nesina treatment.
- 12 months after Nesina treatment: data at 12 months after Nesina treatment will be used for the 12 months survey sheet (electronic) for patients who continued treatment.

For patients who discontinued treatment, data at 12 months after Nesina treatment will not be used for the 12 months survey sheet (electronic).

• 36 months after Nesina treatment: data at 36 months after Nesina treatment will be used for the 36 months survey sheet (electronic) for patients who continued treatment.

For patients who discontinued treatment, data at 36 months after Nesina treatment will not be used for the 36 months survey sheet (electronic).

• At the last evaluation: The last VISIT data within the evaluation period will be used.

## 1.6 Display Data Digit

Display digits are described as below.

| Term | Display digit | Unit |
|---|---|---|
| HbA1c | 0.1 | % |
| Fasting blood glucose level | 1 | mg/dL |
| Fasting insulin level | 0.1 | μU/mL |
| Fasting triglyceride | 1 | mg/dL |
| Total cholesterol | 1 | mg/dL |
| HDL-cholesterol | 1 | mg/dL |
| LDL-cholesterol | 1 | mg/dL |
| Non-HDL cholesterol | 1 | mg/dL |
| Systolic blood pressure | 1 | mmHg |
| Diastolic blood pressure | 1 | mmHg |
| Weight | 0.1 | kg |
| BMI | 0.1 | kg/m <sup>2</sup> |
| Age | 1 | Year |
| Disease duration of type 2 diabetes mellitus | 0.1 | Year |
| Height | 1 | cm |
| Week of pregnancy | 1 | Week |
| Nesina treatment period | 1 | Day |
| Mean daily dose of Nesina | 0.01 | mg |

## 2.0 Disposition of Patients (Patient Diagram)

(1) Patients to be tabulated and analyzed

Registered patients

#### (2) Details of tabulation and analysis

The following will be tabulated: the number of registered patients, number of medical site at which patients is registered, number of patients whose survey sheets (electronic) are collected, number of patients whose survey sheets (electronic) are not collected, number of patients in the Safety Analysis Set, number of patients in the Not Safety Analysis Set, number of patients in the Efficacy Analysis Set, and number of patients in the Not Efficacy Analysis Set.

For the number of medical sites at which patients are registered, do not duplicate the same medical site with different departments.

For patients whose survey sheets (electronic) are not collected, tabulate the number of patients for each reason for not collected survey sheets.

For the Not Safety Analysis Set and Not Efficacy Analysis Set, the number of patients will be tabulated for each reason for exclusion to create the list.

The following is the handling of the decision whether patients who meet the following criteria should be evaluated:

| Criterion | Safety<br>evaluation | Efficacy<br>evaluation |
|---|---|---|
| Pre-agreement administration [found after administration] | × | × |
| Registration 15 days after the start of Nesina treatment [found after registration] | × | × |
| Nesina taking not confirmed [after the end of patient registration period] | × | × |
| No data for post-administration of Nesina | × | × |
| Data reliability was not confirmed | × | × |
| Other than patients with mild type 2 diabetes mellitus | 0 | × |

o Included, × Excluded or not evaluated

#### (3) Number of tables and figures

Figure 2.0-1 and Table 2.0-1

## 3.0 Patient Demographics

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Each parameter will be classified by the categories described below to tabulate the number of patients and frequency.

| Parameter | Category |
|---|---|
| Sex | Male, Female |
| Age | Summary statistics |
| | < 65 years, ≥ 65 years |
| | < 75 years, ≥ 75 years |
| | < 20 years, 20 to 29 years, 30 to 39 years, 40 to 49 years, 50 to 59 years, |
| | 60 to 69 years, 70 to 79 years, $\geq$ 80 years |
| Disease duration of | |
| type 2 diabetes | Summary statistics |
| mellitus | |
| (year) | $<$ 2 years, 2 to $<$ 5 years, 5 to $<$ 10 years, $\ge$ 10 years, Unknown |
| Height | Summary statistics |
| Category of clinical | Outpatient, Inpatient |
| practice | Outpatient, inpatient |
| Pregnancy (only | No, Yes |
| females) | 140, 165 |
| Severity of renal | Normal, Mild, Moderate, Severe |
| impairment | Normal + Mild, Moderate + Severe |
| Concurrent disease | No, Yes |
| Diabetic complication | No, Yes |
| Details of diabetic | Diabetic nephropathy, diabetic retinopathy, diabetic neuropathy |
| complication | For the proportion, the number of patients with diabetic complication |
| (overlapped) | will be denominator. |
| Concurrent | No, Yes |
| hypertension | 140, 165 |
| Concurrent | No, Yes |
| dyslipidemia | 140, 165 |
| Concurrent | No, Yes |
| hyperuricemia | 110, 103 |
| Concurrent liver | No, Yes |
| disorder | 110, 165 |
| Details of concurrent | Hepatic steatosis, alcoholic hepatitis, chronic hepatitis, hepatic |

| Parameter | Category |
|---|---|
| liver disorder | cirrhosis, or other |
| (overlapped) | For the proportion, the number of with concurrent liver disorder will be |
| | denominator. |
| Concurrent renal disorder | No, Yes |
| Details of concurrent renal disorder | Nephrotic syndrome, glomerulonephritis, chronic glomerulonephritis, other For the proportion, the number of with concurrent renal disorder will |
| (overlapped) | be denominator. |
| Concurrent heart disease | No, Yes |
| Details of concurrent | Cardiac failure, myocardial infarction, angina pectoris, other |
| heart disease | For the proportion, the number of with concurrent heart disease will be |
| (overlapped) | denominator. |
| Concurrent cardiac failure | No, Yes |
| Severity classification | Classes NYHA I, NYHA II, NYHA III, and NYHA IV, Unknown |
| of cardiac failure | For the proportion, the number of with concurrent cardiac failure will |
| (NYHA classification) | be denominator. |
| Concurrent stroke-<br>related disease | No, Yes |
| Details of concurrent<br>stroke-related disease<br>(overlapped) | Cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage, transient ischaemic attack For the proportion, the number of with concurrent stroke-related disease will be denominator. |
| Concurrent allergic disease | No, Yes |
| Concurrent malignant tumour | No, Yes |
| Concurrent malignant tumour (narrow sense) | No, Yes |
| Other concurrent disease | No, Yes |
| Past medical history | No, Yes, Unknown |
| Hypersensitivity predisposition | No, Yes, Unknown |
| Alcohol history (drinking alcoholic | Yes, No, Unknown |

| Parameter | Category |
|---|---|
| drinks almost on a | |
| daily basis) | |
| Smoking history | Never, Smoking, Smoked, Unknown |
| HbA1c(NGSP value) | Summary statistics |
| (at the start of Nesina treatment) | $< 6.0\%$ , $6.0\%$ to $< 7.0\%$ , $7.0\%$ to $< 8.0\%$ , $\ge 8.0\%$ , Unknown |
| | ≥7.4%, > 7.4%, Unknown |
| Weight | Summary statistics |
| BMI | Summary statistics |
| | $< 18.5 \text{ kg/m}^2, \ 18.5 \text{ to} < 25 \text{ kg/m}^2, \ 25 \text{ to} < 30 \text{ kg/m}^2, \ge 30 \text{ kg/m}^2,$ |
| | Unknown |
| | $< 25 \text{ kg/m}^2, \ge 25 \text{ kg/m}^2, \text{ Unknown}$ |
| Dietary intervention | |
| (at the start of Nesina | Yes, No |
| treatment) | |
| Exercise intervention | |
| (at the start of Nesina | Yes, No |
| treatment) | |

Table 3.0-1

## 4.0 Details of Treatment

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Each parameter will be classified by the categories described below to tabulate the number of patients and frequency.

| Parameter | Category |
|---|---|
| Initial dose of Nesina | 25 mg, 12.5 mg, 6.25 mg, or other |
| Mean daily dose of<br>Nesina | > 25 mg, 25 to >12.5 mg, 12.5 to > 6.25 mg, or ≤6.25 mg |
| Nesina treatment period | Summary statistics |
| Administration of prior medication (diabetic drug) | No, Yes |
| Prior medications<br>(diabetic drugs) | α-glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, insulin preparations, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, combination of diabetic drugs, or other diabetic drugs For the proportion, the number of patients with "Yes" for administration of prior medication (diabetic drug) will be denominator. |
| Administration of prior medication (other than diabetic drug) | No, Yes |
| Administration of concomitant medication (diabetic drug) | No, Yes |
| Concomitant medications (diabetic drugs) (overlapped) | α-glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, shortrapid-acting insulin secretagogues, insulin preparations, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, combination of diabetic drugs, or other diabetic drugs For the proportion, the number of patients with "Yes" for administration of concomitant medication (diabetic drug) will be denominator. |
| Administration of concomitant medication | No, Yes |

| Parameter | Category |
|---|---|
| (hypertension drug) | |
| Concomitant | ARB, Ca antagonists, ACE inhibitors, diuretics, $\alpha$ blockers, $\alpha\beta/\beta$ |
| medications | blockers, Complication of hypertension drugs, or other |
| (hypertension drugs) | For the proportion, the number of patients with "Yes" for administration |
| (overlapped) | of concomitant medication (hypertension drug) will be denominator. |
| Administration of | |
| concomitant | No, Yes |
| medication | 10, 165 |
| (dyslipidaemia drug) | |
| Concomitant | Statins, fibrates, EPA/DHA, or other |
| medications | For the proportion, the number of patients with "Yes" for administration |
| (dyslipidaemia drugs) | of concomitant medication (dyslipidaemia drug) will be denominator. |
| (overlapped) | of concommant medication (dyshpredefina drug) will be denominator. |
| Administration of | |
| concomitant | No, Yes |
| medication (protease | 1.0, 1.0 |
| drug) | |
| Administration of | |
| concomitant | |
| medication (combined | No, Yes |
| with renal excretory | |
| drug) | |
| Administration of | |
| concomitant | No, Yes |
| medication (other) | |

Table 4.0-1

## 4.1 Initial Dose of Nesina and Mean Daily Dose of Nesina, by Severity of Renal Impairment

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Cross tabulation will be used for the initial dose of Nesina and the mean daily dose of Nesina, by severity of renal impairment.

| Parameter | Category |
|-------------------|--------------------------------|
| Severity of renal | Normal, Mild, Moderate, Severe |
| impairment | Normal, Wild, Woderate, Severe |

| Parameter | Category |
|---|---|
| | Normal + Mild, Moderate + Severe |
| Initial dose of Nesina | 25 mg, 12.5 mg, 6.25 mg, or other |
| Mean daily dose of | > 25 mg, 25 to >12.5 mg, 12.5 to > 6.25 mg, or ≤6.25 mg |
| Nesina | 23 mg, 23 to ≥12.3 mg, 12.3 to ≥ 0.23 mg, or ≤0.23 mg |

Tables 4.1-1 and 4.1-2

## 5.0 Safety Tabulation and Analysis

## 5.1 Occurrence of adverse events and adverse drug reactions / infections

#### 5.1.1 Occurrence of adverse events

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated for adverse events.

Total and mild type 2 diabetes mellitus patients will be tabulated.

| Parameter | Details of analysis |
|---|---|
| Number of patients with adverse events | Number of patients who experienced adverse events. |
| Number of adverse events | Number of adverse events. Count as an event if the same adverse event (LLT) occur multiple times in a patient. Count as different events for different LLTs even if they have the same PT. |
| Percent of patients with adverse events | Described in Section 1.1. |
| Type of adverse events | Will be broadly divided into the SOCs and tabulated by PT in the SOCs. In case of the laboratory test-related events, type of adverse events will be broadly divided into the SOCs and HLGTs for tabulation by PT. For the SOCs, the number of patients with adverse events and percent of patients with events will be described in the order of SOCs agreed internationally. For the PTs, the number of adverse events and percent of events will be described in the ascending order of PT codes. Count as an event if the same adverse event (LLT) occur multiple times in a patient. Count as different events for different LLTs even if they have the same PT. |

## (3) Number of tables and figures

Table 5.1.1-1

## 5.1.2 Occurrence of adverse drug reactions / infections

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated for adverse drug reactions, etc. and serious adverse drug reactions, etc.

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of patients with | |
| adverse drug reactions, | Number of patients who experienced adverse drug reactions, etc. |
| etc. | |
| | Number of adverse drug reactions, etc. Count as an event if the same |
| Number of adverse drug | adverse drug reactions, etc. (LLT) occur multiple times in a patient. |
| reactions, etc. | Count as different events for different LLTs even though they have |
| | the same PT. |
| Percent of patients with | |
| adverse drug reactions, | Described in Section 1.1. |
| etc. | |
| | Will be broadly divided into the SOCs and tabulated by PT in the |
| | SOCs. In case of the laboratory test-related events, type of adverse |
| | events will be broadly divided into the SOCs and HLGTs for |
| | tabulation by PT. |
| | For the SOCs, the number of patients with adverse drug reactions, |
| True of advance days | etc. and percent of patients with adverse drug reactions, etc. will be |
| Type of adverse drug | described in the order of SOCs agreed internationally. |
| reactions, etc. | For the PTs, the number of adverse drug reactions, etc. and percent |
| | of adverse drug reactions, etc. will be described in the ascending |
| | order of PT codes. Count as an event if the same adverse drug |
| | reactions, etc. (LLT) occur multiple times in a patient. Count as |
| | different events for different LLTs even though they have the same |
| | PT. |

Tables 5.1.2-1 and 5.1.2-2

## 5.1.3 Important Identified Risks, Important Potential Risks, and Important Missing Information

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated for important identified risks, important potential risks, and important missing information (described in Section 1.2).

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of patients with<br>adverse events (or<br>adverse drug reactions,<br>etc.) | Number of patients who experienced adverse events (or adverse drug reactions, etc.) with important identified risks, important potential risks, and important missing information. |

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of adverse events (or adverse drug reactions, etc.) | Number of adverse events (or adverse drug reactions, etc.) with important identified risks, important potential risks, and important missing information. Count as an event if the same adverse event (or adverse drug reaction, etc.) (LLT) occur multiple times in a patient. Count as different events for different LLTs even if they have the same PT. |
| Percent of patients with adverse events (or adverse drug reactions, etc.) | Described in Section 1.1. |
| Type of adverse events (or adverse drug reactions, etc.) | Will be broadly divided into the important identified risks, important potential risks, and important missing information and tabulated by PT in them. For the PTs, the number of adverse events (or adverse drug reactions, etc.) and percent of adverse events (or adverse drug reactions, etc.) will be described in the ascending order of PT codes. Count as an event if the same adverse event (or adverse drug reaction, etc.) (LLT) occur multiple times in a patient. Count as different events for different LLTs even though they have the same PT. |

Tables 5.1.3-1 and 5.1.3-2

5.2 Occurrence of Adverse Events and Adverse Drug Reactions / Infections in the Not Safety Analysis

Set

- 5.2.1 Occurrence of Adverse Events
  - (1) Patients to be tabulated and analyzed

Not Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated.

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of patients with adverse events | Number of patients who experienced adverse events. |
| Number of adverse events | Number of adverse events. Count as an event if the same adverse event (LLT) occur multiple times in a patient. |

| Parameter | Details of tabulation and analysis |
|---|---|
| | Count as different events for different LLTs even if they have the |
| | same PT. |
| Percent of patients with | Described in Section 1.1. |
| adverse events | Described in Section 1.1. |
| | Will be broadly divided into the SOCs and tabulated by PT in the |
| | SOCs. In case of the laboratory test-related events, type of adverse |
| | events will be broadly divided into the SOCs and HLGTs for |
| | tabulation by PT. |
| | For the SOCs, the number of patients with adverse events and |
| Type of adverse events | percent of patients with events will be described in the order of |
| Type of adverse events | SOCs agreed internationally. |
| | For the PTs, the number of adverse events and percent of events will |
| | be described in the ascending order of PT codes. Count as an event |
| | if the same adverse event (LLT) occur multiple times in a patient. |
| | Count as different events for different LLTs even though they have |
| | the same PT. |

Table 5.2-1

## 5.2.2 Occurrence of adverse drug reactions / infections

(1) Patients to be tabulated and analyzed

Not Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated.

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of patients with | |
| adverse drug reactions, | Number of patients who experienced adverse drug reactions, etc. |
| etc. | |
| | Number of adverse drug reactions, etc. Count as an event if the same |
| Number of adverse drug | adverse drug reactions, etc. (LLT) occur multiple times in a patient. |
| reactions, etc. | Count as different events for different LLTs even if they have the |
| | same PT. |
| Percent of patients with | |
| adverse drug reactions, | Described in Section 1.1. |
| etc. | |
| Type of adverse drug | Will be broadly divided into the SOCs and tabulated by PT in the |
| reactions, etc. | SOCs. In case of the laboratory test-related events, type of adverse |

| events will be broadly divided into the SOCs and HLGTs for |
|------------------------------------------------------------------------|
| tabulation by PT. |
| For the SOCs, the number of patients with adverse drug reactions, |
| etc. and percent of patients with adverse drug reactions, etc. will be |
| described in the order of SOCs agreed internationally. |
| For the PTs, the number of adverse drug reactions, etc. and percent |
| of adverse drug reactions, etc. will be described in the ascending |
| order of PT codes. Count as an event if the same adverse drug |
| reactions, etc. (LLT) occur multiple times in a patient. Count as |
| different events for different LLTs even though they have the same |
| PT. |

Table 5.2-2

- 5.3 Occurrence of Adverse Drug Reactions / Infections by Severity, Onset Period, and Outcome
  - 5.3.1 Occurrence of Adverse Drug Reactions / Infections by Severity, Onset Period, and Outcome
    - (1) Patients to be tabulated and analyzed Safety Analysis Set
    - (2) Details of tabulation and analysis

Each parameter will be categorized by the categories described below to tabulate the type of adverse drug reactions, etc.

Total and mild type 2 diabetes mellitus patients will be tabulated.

| Parameter | Category |
|---|---|
| Severity | Serious, Not serious |
| Onset period | 1 to 14 days, 15 to 28 days, 29 to 84 days, 85 to 168 days, 169 to |
| | 336 days, 337 to 504 days, 505 to 672 days, 673 to 840 days, 841 to |
| | 1008 days, ≥1009 days, or Unknown |
| Outcome | Resolved, Resolving, Not resolved, Resolved with sequelae, Death, |
| | or Unknown |

The method for tabulation of type adverse drug reactions, etc. is described below:

| Parameter | Details of tabulation and analysis |
|---|---|
| Type of adverse drug reactions, etc. | Will be broadly divided into the SOCs and tabulated by PT in the SOCs. In case of the laboratory test-related events, type of adverse events will be broadly divided into the SOCs and HLGTs for tabulation by PT. For the SOCs, the number of patients with adverse drug reactions, |
| | etc. will be described in the order of SOCs agreed internationally. For the PTs, the number of adverse drug reactions, etc. will be |

| Parameter | Details of tabulation and analysis |
|---|---|
| | described in the ascending order of PT codes. Count as an event if |
| | the same adverse drug reactions, etc. (LLT) occur multiple times in |
| | a patient. Count as different events for different LLTs even if they |
| | have the same PT. However, evaluate an event for the same LLT in |
| | accordance with the following order of priority: |
| | Onset period: earlier event |
| | Severity: Serious → Not serious |
| | Outcome: Death $\rightarrow$ Resolved with Sequelae $\rightarrow$ Not resolved $\rightarrow$ |
| | Resolving $\rightarrow$ Resolved $\rightarrow$ Unknown |

Tables 5.3-1 to 5.3-3

## 5.4 Patient Demographics and Frequency of Adverse Drug Reactions / Infections by Treatment

## 5.4.1 Patients demographics and Frequency of Adverse Drug Reactions / Infections by Treatment

- (1) Patients to be tabulated and analyzed Safety Analysis Set
- (2) Details of tabulation and analysis

Each parameter will be categorized by the categories described below to tabulate the percent of patients with adverse drug reactions, etc.

The Fischer exact test will be used for parameters without rank data. The Mann-Whitney U test will be used for parameters with rank data. (The tests will be used for parameters with asterisk [\*].)

| Parameter | Category |
|---|---|
| Sex* | Male, Female |
| Age* | < 65 years, ≥65 years |
| | < 75 years, ≥75 years |
| Severity of renal impairment* | Normal + Mild, Moderate + Severe |
| Concurrent liver disorder* | No, Yes |
| Concurrent renal disorder* | No, Yes |
| Concurrent heart disease* | No, Yes |
| Details of concurrent heart disease | Cardiac failure, myocardial infarction, or angina pectoris |

| Parameter | Category |
|---|---|
| (overlapped) | |
| Concurrent cardiac failure* | No, Yes |
| Severity classification of cardiac failure (NYHA classification)* | Classes NYHA I, NYHA II, NYHA III, and NYHA IV |
| Concurrent stroke-<br>related disease* | No, Yes |
| Mean daily dose of<br>Nesina | > 25 mg, 25 to >12.5 mg, 12.5 to > 6.25 mg, or ≤6.25 mg |
| Administration of concomitant medication (diabetic drug) | No, Yes |
| Concomitant medications (diabetic drugs) (overlapped) | $\alpha$ -glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, or insulin preparations |
| Administration of concomitant medication (protease drug)* | No, Yes |
| Administration of concomitant medication (combined with renal excretory drug)* | No, Yes |

Table 5.4.1-1

## 5.5 Occurrence of Adverse Drug Reactions / Infections by Age

(1) Patients to be tabulated and analyzed Safety Analysis Set

(2) Details of tabulation and analysis

Age will be classified into < 65 years,  $\ge$ 65 years and < 75 years, and  $\ge$ 75 years for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Tables 5.5-1 to 5.5-2

## 5.6 Occurrence of Adverse Drug Reactions / Infections by Sex

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Sex will be classified into male or female for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.6-1

## 5.7 Occurrence of Adverse Drug Reactions / Infections by Liver Disorder

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent liver disorder will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.7-1

## 5.8 Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Renal Disorder

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent renal disorder will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.8-1

## 5.9 Occurrence of Adverse Drug Reactions / Infections by Severity of Renal Impairment

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Severity of renal impairment will be classified into normal + mild or moderate + severe for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.9-1

## 5.10 Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Heart Disease

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent heart disease will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.10-1

## 5.11 Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Heart Failure

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent heart failure will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

#### Table 5.11-1

## 5.12 Occurrence of Adverse Drug Reactions / Infections by Severity of Heart Failure

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Severity of heart failure will be classified into Class NYHA I, NYHA II, NYHA III, or NYHA IV for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.12-1

## 5.13 Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Stroke-related Disease

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent stroke-related disease will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.13-1

## 5.14 Occurrence of Adverse Drug Reactions / Infections by Mean Daily Dose of Nesina

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

The mean daily dose of Nesina will be classified into > 25 mg, 25 to > 12.5 mg, 12.5 to > 6.25 mg, or  $\le 6.25$  mg for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.14-1

5.15 Occurrence of Adverse Drug Reactions / Infections by Mean Daily Dose of Nesina in Patients with

Special Demographics (Patients with Moderate or Higher Renal Impairment)

(1) Patients to be tabulated and analyzed

Patients with moderate or higher renal impairment in the Safety Analysis Set

(2) Details of tabulation and analysis

The mean daily dose of Nesina will be classified into > 25 mg, 25 to > 12.5 mg, 12.5 to > 6.25 mg, or  $\le 6.25$  mg for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.15-1

5.16 Occurrence of Adverse Drug Reactions / Infections by Administration of Concomitant Medication

(Diabetic Drug)

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Administration of concomitant medication (diabetic drug) will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.16-1

- 5.17 Occurrence of Adverse Drug Reactions / Infections by Concomitant Medication (Diabetic Drug)
  - (1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concomitant medications (diabetic drugs) will be classified into the following drugs:  $\alpha$ -glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, or insulin preparations, for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

#### Table 5.17-1

## 5.18 Occurrence of Adverse Drug Reactions / Infections by Presence of Concomitant Protease Inhibitors

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concomitant protease inhibitor will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.18-1

#### 5.19 Occurrence of Adverse Drug Reactions / Infections by Presence of Concomitant Renal Excretory

Drug

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concomitant renal excretory drug be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.19-1

## 5.20 Change in Laboratory/Measured Data

#### 5.20.1 Vital Signs

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

For blood pressure (systolic/diastolic) and weight, summary statistics will be calculated at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation). For changes from the start of Nesina treatment, summary statistics and the mean 95% confidence intervals will be calculated.
Measured values (mean and standard deviation) of blood pressure (systolic/diastolic) and weight will be plotted. For the changes, the mean changes will be created using a bar graph.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.20.1-1 and Figures 5.20.1-1 to 5.20.1-6

#### 5.20.2 Laboratory Values

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

For laboratory values of fasting triglyceride, total cholesterol, HDL-cholesterol, LDL-cholesterol, and non-HDL cholesterol, summary statistics will be calculated at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation). For changes from the start of Nesina treatment, summary statistics and the mean 95% confidence intervals will be calculated.

The individual laboratory values described above (mean and standard deviation) will be plotted. For the changes, the mean changes will be created using a bar graph.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.20.2-1 and Figures 5.20.2-1 to 5.20.2-10

#### 6.0 Efficacy Tabulation and Analysis

#### 6.1 Changes in HbA1c

(1) Patients to be tabulated and analyzed

Efficacy Analysis Set

(2) Details of tabulation and analysis

For HbA1c (NGSP values), summary statistics will be calculated at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation). For changes, summary statistics and the mean 95% confidence intervals will be calculated and the paired t-test will be performed. Measured values of HbA1c (NGSP values) will be plotted and for the changes a bar graph will be created excluding the unknown category at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina

(3) Number of tables and figures

Table 6.1-1 and Figure 6.1-1

treatment and last evaluation).

#### 6.2 Glycemic control achievement rate (HbA1c)

(1) Patients to be tabulated and analyzed

Efficacy Analysis Set

(2) Details of tabulation and analysis

The Glycemic control achievement rate for HbA1c (NGSP value) will be tabulated (< 7.0%,  $\ge 7.0\%$  / < 6.0%,  $\ge 6.0\%$ ) and a bar graph will be created (< 7.0%,  $\ge 7.0\%$  / < 6.0%,  $\ge 6.0\%$ ) at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation) (the unknown category will be excluded for the bar graph).

(3) Number of tables and figures

Table 6.2-1 and Figure 6.2-1

#### 6.3 Changes in Fasting blood glucose level and Fasting insulin level

(1) Patients to be tabulated and analyzed

Efficacy Analysis Set

(2) Details of tabulation and analysis

For fasting blood glucose level and fasting insulin level, summary statistics will be calculated at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation). For changes, summary statistics and the mean 95% confidence intervals will be calculated and the paired t-test will be performed.

Measured values of fasting blood glucose level and fasting insulin level will be plotted and for

the changes a bar graph will be created excluding the unknown category at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation).

(3) Number of tables and figures

Tables 6.3-1 and 6.3-2 and Figures 6.3-1 and 6.3-2

- 6.4 Changes in HbA1c, etc. by Factor Probably Affecting Efficacy
  - (1) Patients to be tabulated and analyzed

Efficacy Analysis Set

(2) Details of tabulation and analysis

For changes in HbA1c (NGSP values), summary statistics and the mean 95% confidence intervals will be calculated and the paired t-test will be performed at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 24 months, and 36 months after Nesina treatment and last evaluation).

The Glycemic control achievement rate for HbA1c (< 7.0%,  $\ge 7.0\%$  / < 6.0%,  $\ge 6.0\%$ ) at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 24 months, and 36 months after Nesina treatment and last evaluation) will be tabulated at the following parameters:

- i Sex (Male, Female)
- ii Age ( $< 65 \text{ years}, \ge 65 \text{ years}$ )
- iii Age (< 75 years, ≥75 years)
- iv Concurrent renal disorder (No, Yes)
- v HbA1c (NGSP value) at the start of Nesina treatment (< 6.0%, 6.0% to < 7.0%, 7.0% to < 8.0%,  $\geq 8.0\%$ )
- vi Mean daily dose of Nesina (> 25 mg, 25 to > 12.5 mg, 12.5 to > 6.25 mg, or 6.25 mg)
- vii Concomitant diabetic drugs (α-glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, or insulin preparations)
- (3) Number of tables and figures

Tables 6.4-1 to 6.4-14

- 6.5 Changes in HbA1c, etc. in Patients with Special Demographics
  - (1) Patients to be tabulated and analyzed

Efficacy Analysis Set.

However, patients will be evaluated for Parameter (ii) in (2) Details of tabulation and analysis. Patients with moderate or higher renal impairment in the Efficacy Analysis Set.

(2) Details of tabulation and analysis

For changes in HbA1c (NGSP values), summary statistics and the mean 95% confidence intervals will be calculated and the paired t-test will be performed at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 24 months, and 36 months after

Nesina treatment and last evaluation).

The Glycemic control achievement rate for HbA1c ( $< 7.0\%, \ge 7.0\% / < 6.0\%, \ge 6.0\%$ ) at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 24 months, and 36 months after Nesina treatment and last evaluation) will be tabulated at the following parameters:

- i. Severity of renal impairment (Normal + Mild, Moderate + Severe)
- ii. Mean daily dose of Nesina (> 25 mg, 25 to > 12.5 mg, 12.5 to > 6.25 mg, or 6.25 mg)
- (3) Number of tables and figures

Tables 6.5-1 to 6.5-4

# Statistical Analysis Plan

# Nesina Tablets Special Drug Use Surveillance: Mild Type 2 Diabetes Mellitus

(Final Analysis)

Takeda Pharmaceutical Company Limited.

PPD

PPD

Version 2.0, Created on January 30, 2018

## Table of Contents

| 1.0 De | finition of Terms and Handling of Laboratory/Measured Data |
|---|---|
| 1.1 | Definitions |
| 1.2 | Important Identified Risks, Potential Risks, and Missing Information |
| 1.3 | Display digit11 |
| 1.4 | Level of Significance and Confidence Coefficient |
| 1.5 | Handling of Laboratory/Measured Data |
| 1.6 | Display Data Digit |
| 2.0 Dis | sposition of Patients (Patient Diagram)14 |
| 3.0 Pat | ient Demographics |
| 4.0 De | tails of Treatment |
| 4.1 | Initial Dose of Nesina and Mean Daily Dose of Nesina, by Severity of Renal Impairment19 |
| 5.0 Sa | Fety Tabulation and Analysis21 |
| 5.1 | Occurrence of adverse events and adverse drug reactions / infections |
| 5.1.1 | Occurrence of adverse events |
| 5.1.2 | Occurrence of adverse drug reactions / infections |
| 5.1.3 | Important Identified Risks, Important Potential Risks, and Important Missing Information22 |
| 5.2 | Occurrence of Adverse Events and Adverse Drug Reactions / Infections in the Not Safety Analysis |
| Set | 23 |
| 5.2.1 | Occurrence of Adverse Events |
| 5.2.2 | Occurrence of adverse drug reactions / infections |
| 5.3 | Occurrence of Adverse Drug Reactions / Infections by Severity, Onset Period, and Outcome25 |
| 5.3.1 | Occurrence of Adverse Drug Reactions / Infections by Severity, Onset Period, and Outcome 25 |
| 5.4 | Patient Demographics and Frequency of Adverse Drug Reactions / Infections by Treatment26 |
| 5.4.1 | Patients demographics and Frequency of Adverse Drug Reactions / Infections by Treatment .26 |
| 5.5 | Occurrence of Adverse Drug Reactions / Infections by Age |
| 5.6 | Occurrence of Adverse Drug Reactions / Infections by Sex |
| 5.7 | Occurrence of Adverse Drug Reactions / Infections by Liver Disorder |
| 5.8 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Renal Disorder.28 |
| 5.9 | Occurrence of Adverse Drug Reactions / Infections by Severity of Renal Impairment29 |
| 5.10 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Heart Disease29 |
| 5.11 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Heart Failure29 |
| 5.12 | Occurrence of Adverse Drug Reactions / Infections by Severity of Heart Failure30 |
| 5.13 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Stroke-related |
| Disease | 30 |
| 5.14 | Occurrence of Adverse Drug Reactions / Infections by Mean Daily Dose of Nesina30 |
| 5.15 | Occurrence of Adverse Drug Reactions / Infections by Mean Daily Dose of Nesina in Patients with |
| Special | Demographics (Patients with Moderate or Higher Renal Impairment)31 |
| 5.16 | Occurrence of Adverse Drug Reactions / Infections by Administration of Concomitant Medication |

| (Diabeti | c Drug) | 31 |
|---|---|---|
| 5.17 | Occurrence of Adverse Drug Reactions / Infections by Concomitant Medication (Diabeter) | etic Drug) |
| | 31 | |
| 5.18 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concomitant | Protease |
| Inhibito | rs | 32 |
| 5.19 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concomitant Renal | Excretory |
| Drug | 32 | |
| 5.20 | Change in Laboratory/Measured Data | 32 |
| 5.20.1 | Vital Signs | 32 |
| 5.20.2 | Laboratory Values | 33 |
| 6.0 Effi | cacy Tabulation and Analysis | 34 |
| 6.1 | Changes in HbA1c | 34 |
| 6.2 | Glycemic control achievement rate (HbA1c) | 34 |
| 6.3 | Changes in Fasting blood glucose level and Fasting insulin level | 34 |
| 6.4 | Changes in HbA1c, etc. by Factor Probably Affecting Efficacy | 35 |
| 6.5 | Changes in HbA1c, etc. in Patients with Special Demographics | 35 |

# 1.0 Definition of Terms and Handling of Laboratory/Measured Data

# 1.1 Definitions

| Term | Definition |
|---|---|
| Nesina | Nesina tablet(s) is abbreviated as Nesina in this statistical analysis plan. |
| SOC | System Organ Class of MedDRA/J |
| | MedDRA/J version 20.1 is used for this document. |
| HLGT | High level group term of MedDRA/J |
| PT | Preferred term of MedDRA/J |
| LLT | Lowest level term of MedDRA/J |
| Registered patients | Patients whose registration was approved |
| Survey sheet (electronic) | Patients whose survey sheets were sent via |
| collected patients | |
| Survey sheet (electronic) | Of the registered patients, patients whose survey sheets (electronic) were |
| uncollected patients | uncollected. |
| Safety Analysis Set | Of the survey sheet (electronic) collected patients, patients who were |
| | evaluated for safety analysis. |
| | For tabulation, the description of "total" means the Safety Analysis Set. |
| Not Safety Analysis Set | Of the survey sheet (electronic) collected patients, patients who were excluded |
| | from safety analysis |
| Efficacy Analysis Set | Of the Safety Analysis Set, patients who were evaluated for efficacy analysis |
| Not Efficacy Analysis Set | Of the Safety Analysis Set, patients who were excluded from the efficacy |
| | analysis |
| First date of Nesina | Of the start dates of the Nesina treatment period in patients, the earliest date is |
| treatment | defined as the first date of Nesina treatment. |
| Last date of Nesina | Of the last dates of the Nesina treatment period in patients, the latest date is |
| treatment | defined as the last date of Nesina treatment. If Nesina treatment is continued |
| | and the year, month, and date of the continued treatment period are specified, |
| | the year, month, and date of the continued treatment period are defined as the |
| | last date of Nesina treatment. If the data for the year, month, and date of the |
| | continued treatment period are missing, the following date is defined as the |
| | last date of Nesina treatment. |
| | (1) First date of Nesina treatment + 3 years (same month and date), if Nesina |
| | treatment is continued based on the survey sheet (electronic) after 36 |
| | months of treatment* |
| | (2) For other than the above, the first date of Nesina treatment + 1 year (same |
| | month and date), if Nesina treatment is continued based on the survey |
| | sheet (electronic) after 12 months of treatment** |

| Term | Definition |
|---|---|
| | For the continued treatment of Nesina, the following is considered as the "treatment to be continued:" • [End of Nesina tablet treatment] * If "No" for "Did you discontinue Nesina tablets by 12 to 36 months after the start of treatment?" ** If "No" for "Did you discontinue Nesina tablets by 12 months after |
| | the start of treatment?" |
| Adverse drug reactions, etc. | Abbreviation of "adverse drug reactions / infections" Of the adverse events, events for which causal relationship to Nesina was assessed as "Not related" by the Investigator. In this statistical analysis plan, "adverse drug reactions / infections" is used in the headings, while "adverse drug reactions, etc." is used in the sentences and tables. |
| Serious adverse events | Adverse events assessed as "serious" by the Investigator. Events described in the MedDRA coding list in the Takeda Medically Significant AE List will be handled as serious even if the Investigator assesses as "Not serious." |
| Serious adverse drug reactions | Abbreviation of "serious adverse drug reactions / infections" Of the "serious adverse events," the events for which causal relationship to Nesina was assessed as "Not related" by the Investigator |
| Number of patients with events | Number of patients with adverse events or adverse drug reactions, etc. |
| Number of events | Number of adverse events or adverse drug reactions, etc. |
| Percent of patients with events | [For safety analysis calculation in the Safety Analysis Set] The formula is: Number of patients with events / Number of Safety Analysis Set × 100. [For safety analysis calculation in the Not Safety Analysis Set] The formula is: Number of patients with events / Number of Not Safety |
| Percent of events | Analysis Set × 100. [For safety analysis calculation in the Safety Analysis Set] The formula is: Number of events / Number of the Safety Analysis Set × 100. [For safety calculation in the Not Safety Analysis Set] The formula is: Number of events / Number of Not Safety Analysis Set × 100. |
| Onset period | The formula is: Onset date of adverse events (or adverse drug reactions, etc.) – start date of Nesina treatment + 1. |

| Term | Definition |
|---|---|
| | For unknown onset date of adverse events (or adverse drug reactions, etc.), the |
| | onset period will be calculated as 1 day. However, if the start month and date |
| | of Nesina treatment are same as the onset month and date of adverse events |
| | (or adverse drug reactions, etc.), the onset period will be calculated as the start |
| | date of Nesina treatment. |
| Mild type 2 diabetes | Patients who have type 2 diabetes mellitus with HbA1c (NGSP value) of ≤ |
| mellitus | 7.4% at the start date of Nesina treatment |
| Patients with diabetic | Patients with any of the following complications: diabetic nephropathy, |
| complication | diabetic retinopathy, or diabetic neuropathy. |
| Patients with diabetic | Patients with complication of PT Code 10012660 (diabetic end stage renal |
| nephropathy | disease) or 10061835 (diabetic nephropathy). |
| Patients with diabetic | Patients with complication of PT Code 10012688 (diabetic retinal oedema) or |
| retinopathy | 10012689 (diabetic retinopathy). |
| Patients with diabetic | Patients with complication of PT Code 10012645 (diabetic autonomic |
| neuropathy | neuropathy), 10012676 (diabetic mononeuropathy), or 10012680 (diabetic |
| | neuropathy). |
| Patients with concurrent | Patients with concurrent disease of the Standardised MedDRA Query |
| hypertension | (hereinafter SMQ) Code 20000147 (hypertension (SMQ) narrow). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000026 (dyslipidaemia |
| dyslipidemia | (SMQ) narrow). |
| Patients with concurrent | Patients with concurrent disease of the PT code meeting the Takeda MedDRA |
| hyperuricemia | Query 20.1 (hereinafter, TMQ 20.1) (blood uric acid increased). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000005 (hepatic |
| liver disorder | disorders (narrow)). |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10019708 (hepatic steatosis). |
| hepatic steatosis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10019728 (hepatitis |
| alcoholic hepatitis | alcoholic). |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10008909 (chronic hepatitis). |
| chronic hepatitis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10019641 (hepatic cirrhosis). |
| hepatic cirrhosis | |
| Patients with concurrent | Patients with concurrent disease of the TMQ 20.1 (renal disease). |
| renal disorder | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10029164 (nephrotic |
| nephrotic syndrome | syndrome). |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10018364 |
| glomerulonephritis | (glomerulonephritis) or the PT Code 10018367 (glomerulonephritis chronic). |

| Term | Definition |
|---|---|
| Patients with concurrent | Patients with concurrent disease of the PT Code 10064848 (chronic kidney |
| chronic renal failure | disease) or the PT Code 10038435 (renal failure). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10007541 (cardiac |
| heart disease | disorders). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000004 (cardiac failure |
| cardiac failure | (SMQ) narrow). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000047 (myocardial |
| myocardial infarction | infarction (SMQ) narrow). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10007541 (cardiac |
| angina pectoris | disorders) and the PT Code 10036759 (prinzmetal angina), PT Code 10002383 |
| | (angina pectoris), PT Code 10058144 (postinfarction angina), PT Code |
| | 10002388 (angina unstable), or LLT Code 10065566 (microvascular angina). |
| Patients with concurrent | Patients with concurrent disease of cerebral infarction, cerebral haemorrhage, |
| stroke-related disease | subarachnoid haemorrhage, or transient ischaemic attack, described below. |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10006147 (brain stem |
| disease cerebral infarction | infarction), PT Code 10008118 (cerebral infarction), PT Code 10008119 |
| | (cerebral infarction foetal), PT Code 10008034 (cerebellar infarction), PT |
| | Code 10019005 (haemorrhagic cerebral infarction), PT Code 10051078 |
| | (lacunar infarction), PT Code 10056237 (migrainous infarction), PT Code |
| | 10058571 (spinal cord infarction), PT Code 10060839 (embolic cerebral |
| | infarction), PT Code 10060840 (ischaemic cerebral infarction), PT Code |
| | 10064961 (thalamic infarction), PT Code 10067347 (thrombotic cerebral |
| | infarction), or PT Code 10069020 (basal ganglia infarction). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029205 (nervous system |
| cerebral hemorrhage | disorders) and the PT Code 10006145 (brain stem haemorrhage), PT Code |
| | 10008111 (cerebral haemorrhage), PT Code 10008112 (cerebral haemorrhage |
| | neonatal), PT Code 10008030 (cerebellar haemorrhage), PT Code 10018985 |
| | (haemorrhage intracranial), PT Code 10022840 (intraventricular |
| | haemorrhage), PT Code 10022841 (intraventricular haemorrhage neonatal), |
| | PT Code 10042365 (subdural haemorrhage neonatal), PT Code 10049236 |
| | (spinal epidural haemorrhage), PT Code 10048992 (spinal cord haemorrhage), |
| | PT Code 10050157 (cerebral haemorrhage foetal), PT Code 10052593 |
| | (meningorrhagia), PT Code 10058939 (thalamus haemorrhage), PT Code |
| | 10058940 (putamen haemorrhage), PT Code 10067057 (basal ganglia |
| | haemorrhage), PT Code 10067277 (cerebral microhaemorrhage), PT Code |
| | 10071205 (brain stem microhaemorrhage), PT Code 10071206 (cerebellar |
| | microhaemorrhage), PT Code 10072043 (central nervous system |
| | haemorrhage), or PT Code 10073563 (Spinal subdural haemorrhage). |

| Term | Definition |
|---|---|
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029205 (nervous system |
| subarachnoid hemorrhage | disorders) and the PT Code 10042316 (subarachnoid haemorrhage), PT Code |
| | 10042317 (subarachnoid haemorrhage neonatal), PT Code 10073564 (spinal |
| | subarachnoid haemorrhage), LLT Code 10072201 (Asymptomatic |
| | subarachnoid haemorrhage). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029205 (nervous system |
| transient ischemic attack | disorders) and the PT Code 10044390 (transient ischaemic attack). |
| Patients with concurrent | Patients with concurrent disease of bronchial asthma, pollinosis, allergic |
| allergic disease | rhinitis, or allergic dermatitis, described below. |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10038738 (respiratory, |
| bronchial asthma | thoracic and mediastinal disorders) and the PT Code 10003553 (asthma), PT |
| | Code 10075084 (aspirin-exacerbated respiratory disease), PT Code 10003557 |
| | (asthma exercise induced), PT Code 10003559 (asthma late onset), PT Code |
| | 10041961 (status asthmaticus), PT Code 10001890 (alveolitis allergic), PT |
| | Code 10049585 (infantile asthma), PT Code 10070836 (occupational asthma), |
| | or PT Code 10064823 (asthmatic crisis). |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10048908 (seasonal allergy). |
| pollinosis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10039085 (rhinitis allergic). |
| allergic rhinitis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10012434 (dermatitis |
| allergic dermatitis | allergic). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029104 (neoplasms |
| malignant tumor | benign, malignant and unspecified (incl cysts and polyps)). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000194 (malignant |
| malignant tumor (narrow | tumour (SMQ) narrow). |
| sense) | |
| Patients with other | Patients with concurrent disease other than the above (diabetic complication, |
| concurrent disease | hypertension, dyslipidaemia, hyperuricaemia, liver disease, renal disease, |
| | heart disease, stroke-related disease, allergic disease, malignant tumor, or |
| | malignant tumor (narrow sense)). |
| Severity of renal | Severity of renal impairment in the patient demographic section |
| impairment | |

| Term | Definition |
|---|---|
| Age | If the start month and date of Nesina treatment is earlier than the birth month |
| | and date, calculate using the following formula: Start year of Nesina treatment |
| | - birth year $-$ 1. If the birth month and date is earlier than or equal to the start |
| | month and date of Nesina treatment, calculate using the following formula: |
| | Start year of Nesina treatment – birth year. For unknown birth date, the birth |
| | date will be calculated as the 1st day of the birth month. |
| BMI | Calculate using the following formula: Weight (kg) / (0.0001 $\times$ Height (cm) $\times$ |
| | Height (cm)). Indicate to one decimal place rounded from two decimals. |
| Disease duration of type 2 | Calculate using the following formula: (start date of Nesina treatment - |
| diabetes mellitus (year) | diagnosis period of type 2 diabetes mellitus + 1) / 365.25. |
| | For unknown diagnosis month, calculate as January. |
| | Indicate to one decimal place rounded from two decimals. |
| Prior medication | Medications that patients were taking within 3 months before initiation of |
| | Nesina therapy. |
| Concomitant medication | Medications that patients were taking after the start date of Nesina treatment. |
| Start date of other diabetic | Calculate as the start date of survey sheet (electronic). |
| drug and concomitant | |
| medication (other than | |
| diabetic drug) | |
| End date of other diabetic | Calculate as the end date of survey sheet (electronic). |
| drug and concomitant | |
| medication (other than | |
| diabetic drug) | |
| Diabetic drugs | Drugs of the National Health Insurance (NHI) Drug List Code starting with |
| | 3969, 3961, 3962, 2492, 2499410, 2499411, 2499415, or 2499416. |
| α-glucosidase inhibitors | Drugs of the NHI Drug List Code starting with 3969003, 3969004, 3969009, |
| | or 3969102. |
| Thiazolidines | Drugs of the NHI Drug List Code starting with 3969005, 3969007, 3969100, |
| | 3969101, or 3969103. |
| Sulfonylureas | Drugs of the NHI Drug List Code starting with 3961 or 3969101. |
| Biguanides | Drugs of the NHI Drug List Code starting with 3962, 3969100, 3969104, or |
| | 3969105. |
| Rapid-acting insulin | Drugs of the NHI Drug List Code starting with 3969006, 3969008, 3969013, |
| secretagogues | or 3969102. |
| Insulin preparations | Drugs of the NHI Drug List Code starting with 2492. |
| DPP-4 inhibitors | Drugs of the NHI Drug List Code starting with 3969010, 3969011, 3969012, |
| | 3969014, 3969015, 3969016, 3969017, 3969024, 3969025, 3969103, |
| | 3969104, or 3969105. |
| ı | |

| Term | Definition |
|---|---|
| GLP-1 receptor agonists | Drugs of the NHI Drug List Code starting with 2499410, 2499411, 2499415, |
| | or 2499416. |
| SGLT2 inhibitors | Drugs of the NHI Drug List Code starting with 3969018, 3969018, 3969019, |
| | 3969020, 3969021, 3969022, or 3969023. |
| Combination of diabetic | Drugs of the NHI Drug List Code starting with 3969100, 3969101, 3969102, |
| drugs | 3969103, 3969104, or 3969105. |
| Other diabetic drugs | Other diabetic drugs not classified into the above diabetic drug categories ( $\alpha$ - |
| | glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting |
| | insulin secretagogues, insulin preparations, DPP-4 inhibitors, GLP-1 receptor |
| | agonists, SGLT2 inhibitors, or combination of diabetic drugs). |
| Hypertension drugs | ARB Drugs of the NHI Drug List Code starting with the following 7 |
| | numbers: |
| | 2149039, 2149040, 2149041, 2149042, 2149044, 2149046, 2149048, |
| | 2149100, 2149110, 2149111, 2149112, 2149113, 2149114, 2149115, 2149116, |
| | 2149117, 2149118, 2149119, 2149120, 2149121, 2149122 |
| | Ca antagonists Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 2149019, 2149022, 2149027, 2149030, 2149034, 2149035, 2149037, |
| | 2149038, 2149043, 2149400, 2171006, 2171014, 2171019, 2171020, |
| | 2171021, 2171022, 2171405, 2190001, 2149114, 2149115, 2149116, |
| | 2149117, 2149118, 2149120, 2149121, 2149122, 2190101, 2190102, |
| | 2190103, 2190104 |
| | ACE inhibitors Drugs of the NHI Drug List Code starting with the following |
| | 4 numbers: |
| | 2144 |
| | Diuretics Drugs of the NHI Drug List Code starting with numbers 213 or the |
| | following 7 numbers: |
| | 2149003, 2149007, 2149012, 2149110, 2149111, 2149112, 2149113, |
| | 2149119, 2149122<br>α blockers Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 1234400, 214200210, 2149002, 2149015, 2149023, 2149026, 1152, 1149107, |
| | 1149114, 1149115, 2531001, 2149020 |
| | αβ/β blockers Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 2149032, 2149018, 2123014, 2149009, 2123013, 2123003, 2149008, |
| | 2149016, 2442001, 2123011, 2149036, 2123016, 2149700, 2149031, |
| | 2149010, 2123001, 2123F01, 2149029, 2123008, 2149014, 2149021, |

| Term | Definition |
|---|---|
| | 2149028, 2123015, 2123005, 2149025, 2123009, 2123403, 2149033, 2149011 |
| | Complication of hypertension drugs Drugs of the NHI Drug List Code |
| | starting with the following numbers: |
| | 2149110, 2149111, 2149112, 2149113, 2149114, 2149115, 2149116, 2149117, |
| | 2149118, 2149119, 2149120, 2149121, 2149122 |
| | Other Drugs of the NHI Drug List Code starting with the following numbers: |
| | 2149047, 2142004, 2149001, 2149017, 2145 |
| Dyslipidaemia drugs | Statins Drugs of the NHI Drug List Code starting with the following numbers: |
| | 2189010, 2189011, 2189012, 2189013, 2189015, 2189016, 2189017, |
| | 2190101, 2190102, 2190103, 2190104 |
| | Fibrates Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 2183001, 2183002, 2183003, 2183004, 2183005, 2183006 |
| | EPA/DHA Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 2189019, 3399004 |
| | Other Drugs of the NHI Drug List Code starting with the following numbers: |
| | Dugs, other than the above, of the NHI Drug List Code starting with 218, |
| | 2900002, or 3133001. |
| Concomitant medication | Drugs other than the above (diabetic drugs, hypertension drugs, or |
| (other) | dyslipidaemia drugs). |
| Protease Inhibitor | Use the results of the drug name in the survey sheet (electronic) coded with |
| | the NHI Drug List (Appendix 1. List of Protease Inhibitors). |
| Renal excretory drugs | Use the results of the drug name in the survey sheet (electronic) coded with |
| | the NHI Drug List (Appendix 2. List of Renal Excretory Drugs). |
| Nesina treatment period | Actual treatment period from the start date to the end date of Nesina treatment. |
| (days) | However, the washout period is excluded from the treatment period. |
| | Calculate using the following formula: End of Nesina treatment – start date of |
| | Nesina treatment + 1 (grand total). |
| | (Consider the washout period.) |
| Mean daily dose of Nesina | Calculate using the following formula: Total of "daily dose of Nesina × Nesina |
| | treatment period at the relevant dose" / Nesina treatment period. For the |
| | calculation of Nesina treatment period, refer to the above. |
| | If the daily dose of Nesina is a number outside specification in the survey sheet |
| | (electronic) and is actual number, use the relevant number. |

| Term | Definition |
|---|---|
| HbA1c (NGSP value) | The NGSP value only will be used in this analysis. |
| | For the HbA1c (JDS value), calculate using the following formula: |
| | NGSP value (%) = $1.02 \times JDS$ value (%) + $0.25\%$ |
| | The HbA1c (international standard value) will be handled as the NGSP value. |
| Change in HbA1c | For HbA1c converted to the NGSP value, calculate using the following |
| | formula: Laboratory value at each testing time point - Laboratory value at the |
| | start of Nesina treatment. |
| Glycemic control | Divide the following two categories for the Glycemic control achievement |
| achievement rate | rate: |
| | HbA1c (NGSP converted value) [Unit %] |
| | NGSP (%): < 6.0, ≥6.0 / < 7.0,≥ 7.0 |
| non-HDL cholesterol | Calculate using the following formula: "Total cholesterol" - "HDL |
| | cholesterol." |
| Summary statistics | Number of patients, mean, standard deviation, minimum, first quartile, |
| | median, third quartile, and maximum. |

## 1.2 Important Identified Risks, Potential Risks, and Missing Information

| Term | Definition |
|---|---|
| Important identified risk | |
| Hypoglycemia | Adverse events of the following PT Codes (term) are defined as hypoglycemia. |
| | 10020994(Hypoglycaemia neonatal) |
| | 10040576(Shock hypoglycaemic) |
| | 10021000(Hypoglycaemic coma) |
| | 10020993(Hypoglycaemia) |
| | 10065981(Hypoglycaemic unconsciousness) |
| | 10021002(Hypoglycaemic encephalopathy) |
| | 10048803(Hypoglycaemic seizure) |
| | 10020997(Hypoglycaemia unawareness) |
| | 10077216(Hyperinsulinaemic hypoglycaemia) |
| | 10059035(Postprandial hypoglycaemia) |
| Acute pancreatitis | Adverse events of the SMQ Code 20000022 (acute pancreatitis (SMQ) narrow |
| | scope are defined as acute pancreatitis. |
| Hepatic impairment / | Adverse events of the SMQ Code 20000005 (hepatic disorders (SMQ) broad) |
| jaundice | are defined as hepatic impairment / jaundice. |
| Skin disorder including | Adverse events of the SMQ Code 20000020 (severe skin adverse reactions |
| oculomucocutaneous | (SMQ) narrow) are defined as skin disorder including oculomucocutaneous |
| syndrome (Stevens- | syndrome (Stevens-Johnson syndrome) / erythema multiforme. |
| Johnson syndrome) / | |
| erythema multiforme | |
| Rhabdomyolysis | Adverse events of the SMQ Code 20000002 (rhabdomyolysis/myopathy |
| | (SMQ) narrow) are defined as rhabdomyolysis. |
| Intestinal obstruction | Adverse events of the SMQ Code 20000105 (gastrointestinal obstruction |
| | (SMQ) narrow) or the HLGT Code 10018008 (gastrointestinal stenosis and |
| | obstruction) or HLT Code 10052736 (non-mechanical ileus) are defined as |
| | intestinal obstruction. |
| Interstitial pneumonia | Adverse events of the SMQ Code 20000042 (interstitial lung disease (SMQ) |
| | narrow) are defined as interstitial pneumonia. |
| Angioedema | Adverse events of the SMQ Code 20000024 (angioedema (SMQ) narrow) are |
| | defined as angioedema. |
| Important potential risk | |
| Infection | Adverse events of SOC Code 10021881(infections and infestations) are |
| | defined as infection. |
| Malignant tumor | Adverse events of the SOC Code 10029104 (neoplasms benign, malignant |
| | and unspecified (incl cysts and polyps)) are defined as malignant tumor. |
| Malignant tumor (narrow | Adverse events of the SMQ Code 20000194 (malignant tumors (SMQ) |

| Term | Definition |
|---|---|
| sense) | narrow) are defined as malignant tumor (narrow sense). |
| Pemphigoid | Adverse events of the PT Code 10067776 (ocular pemphigoid) or 10034277 |
| | (pemphigoid) are defined as pemphigoid. |

| Term | Definition |
|---|---|
| Important missing | |
| information | |
| Cardiovascular system risk | Adverse events of the SMQ Code 20000047 (myocardial infarction (SMQ) |
| | broad) or SMQ Code 20000061 (central nervous system haemorrhages and |
| | cerebrovascular conditions (SMQ) broad) are defined as cardiovascular |
| | system risk. |
| | "Central nervous system haemorrhage and cerebrovascular conditions (SMQ) |
| | broad" includes the following SMQ classes. |
| | > 20000166(Conditions associated with central nervous system |
| | haemorrhages and cerebrovascular accidents (SMQ) broad) |
| | > 20000064(Cerebrovascular disorder haemorrhagic (SMQ) |
| | broad) |
| | > 20000063(Cerebrovascular disease ischaemic (SMQ) broad) |

# 1.3 Display digit

| Term | Definition |
|---|---|
| Percentage (%) | Percent of patients with adverse events or adverse drug reactions, etc. or percent |
| | of adverse events or adverse drug reactions, etc.: |
| | Indicate to two decimal places rounded from three decimals. |
| | Other than the above: |
| | Indicate to one decimal place rounded from two decimals. |
| Summary statistics | Mean, median, first quartile, and third quartile: |
| | Indicate one lower digit rounded from two lower digits than the digit of the |
| | to-be evaluated data. |
| | Standard deviation: |
| | Indicate two lower digits rounded from three lower digits of the to-be |
| | evaluated data. |
| | Minimum and maximum |
| | Indicate the same digit number as that of the to-be evaluated data (refer to |
| | <u>Section 1.6</u> ). |
| p-value | Indicate to three decimal places rounded down from four decimals. |

| Term | Definition |
|---|---|
| | If the data is rounded down from four decimal places and less than 0.001, display |
| | as $p < 0.001$ . |

#### 1.4 Level of Significance and Confidence Coefficient

Two-sided 5%, two-sided 95%.

#### 1.5 Handling of Laboratory/Measured Data

- VISIT as described in the survey sheet will be used for data other than 12 months and 36 months after Nesina treatment.
- 12 months after Nesina treatment: data at 12 months after Nesina treatment will be used for the 12 months survey sheet (electronic) for patients who continued treatment.

For patients who discontinued treatment, data at 12 months after Nesina treatment will not be used for the 12 months survey sheet (electronic).

• 36 months after Nesina treatment: data at 36 months after Nesina treatment will be used for the 36 months survey sheet (electronic) for patients who continued treatment.

For patients who discontinued treatment, data at 36 months after Nesina treatment will not be used for the 36 months survey sheet (electronic).

• At the last evaluation: The last VISIT data within the evaluation period will be used.

#### 1.6 Display Data Digit

Display digits are described as below.

| Term | Display digit | Unit |
|---|---|---|
| HbA1c | 0.1 | % |
| Fasting blood glucose level | 1 | mg/dL |
| Fasting insulin level | 0.1 | μU/mL |
| Fasting triglyceride | 1 | mg/dL |
| Total cholesterol | 1 | mg/dL |
| HDL-cholesterol | 1 | mg/dL |
| LDL-cholesterol | 1 | mg/dL |
| Non-HDL cholesterol | 1 | mg/dL |
| Systolic blood pressure | 1 | mmHg |
| Diastolic blood pressure | 1 | mmHg |
| Weight | 0.1 | kg |
| BMI | 0.1 | kg/m <sup>2</sup> |
| Age | 1 | Year |
| Disease duration of type 2 diabetes mellitus | 0.1 | Year |
| Height | 1 | cm |
| Week of pregnancy | 1 | Week |
| Nesina treatment period | 1 | Day |
| Mean daily dose of Nesina | 0.01 | mg |

#### 2.0 Disposition of Patients (Patient Diagram)

(1) Patients to be tabulated and analyzed

Registered patients

#### (2) Details of tabulation and analysis

The following will be tabulated: the number of registered patients, number of medical site at which patients is registered, number of patients whose survey sheets (electronic) are collected, number of patients whose survey sheets (electronic) are not collected, number of patients in the Safety Analysis Set, number of patients in the Not Safety Analysis Set, number of patients in the Efficacy Analysis Set, and number of patients in the Not Efficacy Analysis Set.

For the number of medical sites at which patients are registered, do not duplicate the same medical site with different departments.

For patients whose survey sheets (electronic) are not collected, tabulate the number of patients for each reason for not collected survey sheets.

For the Not Safety Analysis Set and Not Efficacy Analysis Set, the number of patients will be tabulated for each reason for exclusion to create the list.

The following is the handling of the decision whether patients who meet the following criteria should be evaluated:

| Criterion | Safety<br>evaluation | Efficacy<br>evaluation |
|---|---|---|
| Pre-agreement administration [found after administration] | × | × |
| Registration 15 days after the start of Nesina treatment [found after registration] | × | × |
| Nesina taking not confirmed [after the end of patient registration period] | × | × |
| No data for post-administration of Nesina | × | × |
| Other than patients with mild type 2 diabetes mellitus | 0 | × |

o Included, × Excluded or not evaluated

#### (3) Number of tables and figures

Figure 2.0-1 and Table 2.0-1

## 3.0 Patient Demographics

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Each parameter will be classified by the categories described below to tabulate the number of patients and frequency.

| Parameter | Category |
|---|---|
| Sex | Male, Female |
| Age | Summary statistics |
| | < 65 years, ≥ 65 years |
| | < 75 years, ≥ 75 years |
| | < 20 years, 20 to 29 years, 30 to 39 years, 40 to 49 years, 50 to 59 years, |
| | 60 to 69 years, 70 to 79 years, $\geq$ 80 years |
| Disease duration of | |
| type 2 diabetes | Summary statistics |
| mellitus | |
| (year) | $<$ 2 years, 2 to $<$ 5 years, 5 to $<$ 10 years, $\ge$ 10 years, Unknown |
| Height | Summary statistics |
| Category of clinical | Outpatient, Inpatient |
| practice | Outpatient, inpatient |
| Pregnancy (only | No, Yes |
| females) | 140, 165 |
| Severity of renal | Normal, Mild, Moderate, Severe |
| impairment | Normal + Mild, Moderate + Severe |
| Concurrent disease | No, Yes |
| Diabetic complication | No, Yes |
| Details of diabetic | Diabetic nephropathy, diabetic retinopathy, diabetic neuropathy |
| complication | For the proportion, the number of patients with diabetic complication |
| (overlapped) | will be denominator. |
| Concurrent | No, Yes |
| hypertension | 140, 165 |
| Concurrent | No, Yes |
| dyslipidemia | 140, 165 |
| Concurrent | No, Yes |
| hyperuricemia | 110, 103 |
| Concurrent liver | No, Yes |
| disorder | 110, 165 |
| Details of concurrent | Hepatic steatosis, alcoholic hepatitis, chronic hepatitis, hepatic |

| Parameter | Category |
|---|---|
| liver disorder | cirrhosis, or other |
| (overlapped) | For the proportion, the number of with concurrent liver disorder will be |
| | denominator. |
| Concurrent renal disorder | No, Yes |
| Details of concurrent renal disorder | Nephrotic syndrome, glomerulonephritis, chronic glomerulonephritis, other For the proportion, the number of with concurrent renal disorder will |
| (overlapped) | be denominator. |
| Concurrent heart disease | No, Yes |
| Details of concurrent | Cardiac failure, myocardial infarction, angina pectoris, other |
| heart disease | For the proportion, the number of with concurrent heart disease will be |
| (overlapped) | denominator. |
| Concurrent cardiac failure | No, Yes |
| Severity classification | Classes NYHA I, NYHA II, NYHA III, and NYHA IV, Unknown |
| of cardiac failure | For the proportion, the number of with concurrent cardiac failure will |
| (NYHA classification) | be denominator. |
| Concurrent stroke-<br>related disease | No, Yes |
| Details of concurrent<br>stroke-related disease<br>(overlapped) | Cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage, transient ischaemic attack For the proportion, the number of with concurrent stroke-related disease will be denominator. |
| Concurrent allergic disease | No, Yes |
| Concurrent malignant tumour | No, Yes |
| Concurrent malignant tumour (narrow sense) | No, Yes |
| Other concurrent disease | No, Yes |
| Past medical history | No, Yes, Unknown |
| Hypersensitivity predisposition | No, Yes, Unknown |
| Alcohol history (drinking alcoholic | Yes, No, Unknown |

| Parameter | Category |
|---|---|
| drinks almost on a | |
| daily basis) | |
| Smoking history | Never, Smoking, Smoked, Unknown |
| HbA1c(NGSP value) | Summary statistics |
| (at the start of Nesina treatment) | $< 6.0\%$ , $6.0\%$ to $< 7.0\%$ , $7.0\%$ to $< 8.0\%$ , $\ge 8.0\%$ , Unknown |
| | ≥7.4%, > 7.4%, Unknown |
| Weight | Summary statistics |
| BMI | Summary statistics |
| | $< 18.5 \text{ kg/m}^2, \ 18.5 \text{ to} < 25 \text{ kg/m}^2, \ 25 \text{ to} < 30 \text{ kg/m}^2, \ge 30 \text{ kg/m}^2,$ |
| | Unknown |
| | $< 25 \text{ kg/m}^2, \ge 25 \text{ kg/m}^2, \text{ Unknown}$ |
| Dietary intervention | |
| (at the start of Nesina | Yes, No |
| treatment) | |
| Exercise intervention | |
| (at the start of Nesina | Yes, No |
| treatment) | |

Table 3.0-1

#### 4.0 Details of Treatment

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Each parameter will be classified by the categories described below to tabulate the number of patients and frequency.

| Parameter | Category |
|---|---|
| Initial dose of Nesina | 25 mg, 12.5 mg, 6.25 mg, or other |
| Mean daily dose of<br>Nesina | > 25 mg, 25 to >12.5 mg, 12.5 to > 6.25 mg, or ≤6.25 mg |
| Nesina treatment period | Summary statistics |
| Administration of prior medication (diabetic drug) | No, Yes |
| Prior medications<br>(diabetic drugs) | α-glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, insulin preparations, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, combination of diabetic drugs, or other diabetic drugs For the proportion, the number of patients with "Yes" for administration of prior medication (diabetic drug) will be denominator. |
| Administration of prior medication (other than diabetic drug) | No, Yes |
| Administration of concomitant medication (diabetic drug) | No, Yes |
| Concomitant medications (diabetic drugs) (overlapped) | α-glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, insulin preparations, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, combination of diabetic drugs, or other diabetic drugs For the proportion, the number of patients with "Yes" for administration of concomitant medication (diabetic drug) will be denominator. |
| Administration of concomitant medication | No, Yes |

| Parameter | Category |
|---|---|
| (hypertension drug) | |
| Concomitant | ARB, Ca antagonists, ACE inhibitors, diuretics, $\alpha$ blockers, $\alpha\beta/\beta$ |
| medications | blockers, Complication of hypertension drugs, or other |
| (hypertension drugs) | For the proportion, the number of patients with "Yes" for administration |
| (overlapped) | of concomitant medication (hypertension drug) will be denominator. |
| Administration of | |
| concomitant | No, Yes |
| medication | 10, 165 |
| (dyslipidaemia drug) | |
| Concomitant | Statins, fibrates, EPA/DHA, or other |
| medications | For the proportion, the number of patients with "Yes" for administration |
| (dyslipidaemia drugs) | of concomitant medication (dyslipidaemia drug) will be denominator. |
| (overlapped) | of concommant medication (dyshpredefina drug) will be denominator. |
| Administration of | |
| concomitant | No, Yes |
| medication (protease | 1.0, 1.0 |
| drug) | |
| Administration of | |
| concomitant | |
| medication (combined | No, Yes |
| with renal excretory | |
| drug) | |
| Administration of | |
| concomitant | No, Yes |
| medication (other) | |

Table 4.0-1

## 4.1 Initial Dose of Nesina and Mean Daily Dose of Nesina, by Severity of Renal Impairment

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Cross tabulation will be used for the initial dose of Nesina and the mean daily dose of Nesina, by severity of renal impairment.

| Parameter | | Category |
|----------------|------|---------------------------------|
| Severity of re | enal | Normal, Mild, Moderate, Severe |
| impairment | | Normai, wind, wioderate, Severe |

| Parameter | Category |
|---|---|
| | Normal + Mild, Moderate + Severe |
| Initial dose of Nesina | 25 mg, 12.5 mg, 6.25 mg, or other |
| Mean daily dose of | 25 25 25 20 5 20 5 20 5 20 5 20 5 20 5 |
| Nesina | $>$ 25 mg, 25 to $>$ 12.5 mg, 12.5 to $>$ 6.25 mg, or $\le$ 6.25 mg |

Tables 4.1-1 and 4.1-2

#### 5.0 Safety Tabulation and Analysis

#### 5.1 Occurrence of adverse events and adverse drug reactions / infections

#### 5.1.1 Occurrence of adverse events

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated for adverse events.

Total and mild type 2 diabetes mellitus patients will be tabulated.

| Parameter | Details of analysis |
|---|---|
| Number of patients with adverse events | Number of patients who experienced adverse events. |
| Number of adverse events | Number of adverse events. Count as an event if the same adverse event (LLT) occur multiple times in a patient. Count as different events for different LLTs even if they have the same PT. |
| Percent of patients with adverse events | Described in Section 1.1. |
| Type of adverse events | Will be broadly divided into the SOCs and tabulated by PT in the SOCs. In case of the laboratory test-related events, type of adverse events will be broadly divided into the SOCs and HLGTs for tabulation by PT. For the SOCs, the number of patients with adverse events and percent of patients with events will be described in the order of SOCs agreed internationally. For the PTs, the number of adverse events and percent of events will be described in the ascending order of PT codes. Count as an event if the same adverse event (LLT) occur multiple times in a patient. Count as different events for different LLTs even if they have the same PT. |

#### (3) Number of tables and figures

Table 5.1.1-1

#### 5.1.2 Occurrence of adverse drug reactions / infections

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated for adverse drug reactions, etc. and serious adverse drug reactions, etc.

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of patients with | |
| adverse drug reactions, | Number of patients who experienced adverse drug reactions, etc. |
| etc. | |
| | Number of adverse drug reactions, etc. Count as an event if the same |
| Number of adverse drug | adverse drug reactions, etc. (LLT) occur multiple times in a patient. |
| reactions, etc. | Count as different events for different LLTs even though they have |
| | the same PT. |
| Percent of patients with | |
| adverse drug reactions, | Described in Section 1.1. |
| etc. | |
| | Will be broadly divided into the SOCs and tabulated by PT in the |
| | SOCs. In case of the laboratory test-related events, type of adverse |
| | events will be broadly divided into the SOCs and HLGTs for |
| | tabulation by PT. |
| | For the SOCs, the number of patients with adverse drug reactions, |
| True of advance days | etc. and percent of patients with adverse drug reactions, etc. will be |
| Type of adverse drug | described in the order of SOCs agreed internationally. |
| reactions, etc. | For the PTs, the number of adverse drug reactions, etc. and percent |
| | of adverse drug reactions, etc. will be described in the ascending |
| | order of PT codes. Count as an event if the same adverse drug |
| | reactions, etc. (LLT) occur multiple times in a patient. Count as |
| | different events for different LLTs even though they have the same |
| | PT. |

Tables 5.1.2-1 and 5.1.2-2

#### 5.1.3 Important Identified Risks, Important Potential Risks, and Important Missing Information

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated for important identified risks, important potential risks, and important missing information (described in Section 1.2).

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of patients with<br>adverse events (or<br>adverse drug reactions,<br>etc.) | Number of patients who experienced adverse events (or adverse drug reactions, etc.) with important identified risks, important potential risks, and important missing information. |

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of adverse events<br>(or adverse drug<br>reactions, etc.) | Number of adverse events (or adverse drug reactions, etc.) with important identified risks, important potential risks, and important missing information. Count as an event if the same adverse event (or adverse drug reaction, etc.) (LLT) occur multiple times in a patient. Count as different events for different LLTs even if they have the same PT. |
| Percent of patients with adverse events (or adverse drug reactions, etc.) | Described in Section 1.1. |
| Type of adverse events (or adverse drug reactions, etc.) | Will be broadly divided into the important identified risks, important potential risks, and important missing information and tabulated by PT in them. For the PTs, the number of adverse events (or adverse drug reactions, etc.) and percent of adverse events (or adverse drug reactions, etc.) will be described in the ascending order of PT codes. Count as an event if the same adverse event (or adverse drug reaction, etc.) (LLT) occur multiple times in a patient. Count as different events for different LLTs even though they have the same PT. |

Tables 5.1.3-1 and 5.1.3-2

5.2 Occurrence of Adverse Events and Adverse Drug Reactions / Infections in the Not Safety Analysis

Set

- 5.2.1 Occurrence of Adverse Events
  - (1) Patients to be tabulated and analyzed

Not Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated.

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of patients with adverse events | Number of patients who experienced adverse events. |
| Number of adverse events | Number of adverse events. Count as an event if the same adverse event (LLT) occur multiple times in a patient. |

| Parameter | Details of tabulation and analysis |
|---|---|
| | Count as different events for different LLTs even if they have the |
| | same PT. |
| Percent of patients with | Described in Section 1.1. |
| adverse events | Described in Section 1.1. |
| | Will be broadly divided into the SOCs and tabulated by PT in the |
| | SOCs. In case of the laboratory test-related events, type of adverse |
| | events will be broadly divided into the SOCs and HLGTs for |
| | tabulation by PT. |
| | For the SOCs, the number of patients with adverse events and |
| Type of adverse events | percent of patients with events will be described in the order of |
| Type of adverse events | SOCs agreed internationally. |
| | For the PTs, the number of adverse events and percent of events will |
| | be described in the ascending order of PT codes. Count as an event |
| | if the same adverse event (LLT) occur multiple times in a patient. |
| | Count as different events for different LLTs even though they have |
| | the same PT. |

Table 5.2-1

#### 5.2.2 Occurrence of adverse drug reactions / infections

(1) Patients to be tabulated and analyzed

Not Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated.

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of patients with | |
| adverse drug reactions, | Number of patients who experienced adverse drug reactions, etc. |
| etc. | |
| | Number of adverse drug reactions, etc. Count as an event if the same |
| Number of adverse drug | adverse drug reactions, etc. (LLT) occur multiple times in a patient. |
| reactions, etc. | Count as different events for different LLTs even if they have the |
| | same PT. |
| Percent of patients with | |
| adverse drug reactions, | Described in Section 1.1. |
| etc. | |
| Type of adverse drug | Will be broadly divided into the SOCs and tabulated by PT in the |
| reactions, etc. | SOCs. In case of the laboratory test-related events, type of adverse |

| events will be broadly divided into the SOCs and HLGTs for |
|------------------------------------------------------------------------|
| tabulation by PT. |
| For the SOCs, the number of patients with adverse drug reactions, |
| etc. and percent of patients with adverse drug reactions, etc. will be |
| described in the order of SOCs agreed internationally. |
| For the PTs, the number of adverse drug reactions, etc. and percent |
| of adverse drug reactions, etc. will be described in the ascending |
| order of PT codes. Count as an event if the same adverse drug |
| reactions, etc. (LLT) occur multiple times in a patient. Count as |
| different events for different LLTs even though they have the same |
| PT. |

Table 5.2-2

- 5.3 Occurrence of Adverse Drug Reactions / Infections by Severity, Onset Period, and Outcome
  - 5.3.1 Occurrence of Adverse Drug Reactions / Infections by Severity, Onset Period, and Outcome
    - (1) Patients to be tabulated and analyzed Safety Analysis Set
    - (2) Details of tabulation and analysis

Each parameter will be categorized by the categories described below to tabulate the type of adverse drug reactions, etc.

Total and mild type 2 diabetes mellitus patients will be tabulated.

| Parameter | Category |
|---|---|
| Severity | Serious, Not serious |
| Onset period | 1 to 14 days, 15 to 28 days, 29 to 84 days, 85 to 168 days, 169 to |
| | 336 days, 337 to 504 days, 505 to 672 days, 673 to 840 days, 841 to |
| | 1008 days, ≥1009 days, or Unknown |
| Outcome | Resolved, Resolving, Not resolved, Resolved with sequelae, Death, |
| | or Unknown |

The method for tabulation of type adverse drug reactions, etc. is described below:

| Parameter | Details of tabulation and analysis |
|---|---|
| Type of adverse drug reactions, etc. | Will be broadly divided into the SOCs and tabulated by PT in the SOCs. In case of the laboratory test-related events, type of adverse events will be broadly divided into the SOCs and HLGTs for tabulation by PT. For the SOCs, the number of patients with adverse drug reactions, |
| | etc. will be described in the order of SOCs agreed internationally. For the PTs, the number of adverse drug reactions, etc. will be |

| Parameter | Details of tabulation and analysis |
|---|---|
| | described in the ascending order of PT codes. Count as an event if |
| | the same adverse drug reactions, etc. (LLT) occur multiple times in |
| | a patient. Count as different events for different LLTs even if they |
| | have the same PT. However, evaluate an event for the same LLT in |
| | accordance with the following order of priority: |
| | Onset period: earlier event |
| | Severity: Serious → Not serious |
| | Outcome: Death $\rightarrow$ Resolved with Sequelae $\rightarrow$ Not resolved $\rightarrow$ |
| | Resolving $\rightarrow$ Resolved $\rightarrow$ Unknown |

Tables 5.3-1 to 5.3-3

#### 5.4 Patient Demographics and Frequency of Adverse Drug Reactions / Infections by Treatment

#### 5.4.1 Patients demographics and Frequency of Adverse Drug Reactions / Infections by Treatment

- (1) Patients to be tabulated and analyzed Safety Analysis Set
- (2) Details of tabulation and analysis

Each parameter will be categorized by the categories described below to tabulate the percent of patients with adverse drug reactions, etc.

The Fischer exact test will be used for parameters without rank data. The Mann-Whitney U test will be used for parameters with rank data. (The tests will be used for parameters with asterisk [\*].)

| Parameter | Category |
|---|---|
| Sex* | Male, Female |
| Age* | < 65 years, ≥65 years |
| | < 75 years, ≥75 years |
| Severity of renal impairment* | Normal + Mild, Moderate + Severe |
| Concurrent liver disorder* | No, Yes |
| Concurrent renal disorder* | No, Yes |
| Concurrent heart disease* | No, Yes |
| Details of concurrent heart disease | Cardiac failure, myocardial infarction, or angina pectoris |

| Parameter | Category |
|---|---|
| (overlapped) | |
| Concurrent cardiac failure* | No, Yes |
| Severity classification of cardiac failure (NYHA classification)* | Classes NYHA I, NYHA II, NYHA III, and NYHA IV |
| Concurrent stroke-<br>related disease* | No, Yes |
| Mean daily dose of<br>Nesina | > 25 mg, 25 to >12.5 mg, 12.5 to > 6.25 mg, or ≤6.25 mg |
| Administration of concomitant medication (diabetic drug) | No, Yes |
| Concomitant medications (diabetic drugs) (overlapped) | $\alpha$ -glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, or insulin preparations |
| Administration of concomitant medication (protease drug)* | No, Yes |
| Administration of concomitant medication (combined with renal excretory drug)* | No, Yes |

Table 5.4.1-1

## 5.5 Occurrence of Adverse Drug Reactions / Infections by Age

(1) Patients to be tabulated and analyzed Safety Analysis Set

(2) Details of tabulation and analysis

Age will be classified into < 65 years,  $\ge$ 65 years and < 75 years, and  $\ge$ 75 years for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Tables 5.5-1 to 5.5-2

#### 5.6 Occurrence of Adverse Drug Reactions / Infections by Sex

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Sex will be classified into male or female for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.6-1

#### 5.7 Occurrence of Adverse Drug Reactions / Infections by Liver Disorder

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent liver disorder will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.7-1

#### 5.8 Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Renal Disorder

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent renal disorder will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.8-1

#### 5.9 Occurrence of Adverse Drug Reactions / Infections by Severity of Renal Impairment

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Severity of renal impairment will be classified into normal + mild or moderate + severe for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.9-1

#### 5.10 Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Heart Disease

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent heart disease will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.10-1

#### 5.11 Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Heart Failure

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent heart failure will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures
#### Table 5.11-1

# 5.12 Occurrence of Adverse Drug Reactions / Infections by Severity of Heart Failure

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Severity of heart failure will be classified into Class NYHA I, NYHA II, NYHA III, or NYHA IV for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.12-1

# 5.13 Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Stroke-related Disease

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent stroke-related disease will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.13-1

# 5.14 Occurrence of Adverse Drug Reactions / Infections by Mean Daily Dose of Nesina

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

The mean daily dose of Nesina will be classified into > 25 mg, 25 to > 12.5 mg, 12.5 to > 6.25 mg, or  $\le 6.25$  mg for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.14-1

5.15 Occurrence of Adverse Drug Reactions / Infections by Mean Daily Dose of Nesina in Patients with

Special Demographics (Patients with Moderate or Higher Renal Impairment)

(1) Patients to be tabulated and analyzed

Patients with moderate or higher renal impairment in the Safety Analysis Set

(2) Details of tabulation and analysis

The mean daily dose of Nesina will be classified into > 25 mg, 25 to > 12.5 mg, 12.5 to > 6.25 mg, or  $\le 6.25$  mg for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.15-1

5.16 Occurrence of Adverse Drug Reactions / Infections by Administration of Concomitant Medication

(Diabetic Drug)

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Administration of concomitant medication (diabetic drug) will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.16-1

- 5.17 Occurrence of Adverse Drug Reactions / Infections by Concomitant Medication (Diabetic Drug)
  - (1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concomitant medications (diabetic drugs) will be classified into the following drugs:  $\alpha$ -glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, or insulin preparations, for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

#### Table 5.17-1

# 5.18 Occurrence of Adverse Drug Reactions / Infections by Presence of Concomitant Protease Inhibitors

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concomitant protease inhibitor will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.18-1

### 5.19 Occurrence of Adverse Drug Reactions / Infections by Presence of Concomitant Renal Excretory

Drug

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concomitant renal excretory drug be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.19-1

# 5.20 Change in Laboratory/Measured Data

#### 5.20.1 Vital Signs

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

For blood pressure (systolic/diastolic) and weight, summary statistics will be calculated at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation). For changes from the start of Nesina treatment, summary statistics and the mean 95% confidence intervals will be calculated.

Measured values (mean and standard deviation) of blood pressure (systolic/diastolic) and weight will be plotted. For the changes, the mean changes will be created using a bar graph.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.20.1-1 and Figures 5.20.1-1 to 5.20.1-6

#### 5.20.2 Laboratory Values

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

For laboratory values of fasting triglyceride, total cholesterol, HDL-cholesterol, LDL-cholesterol, and non-HDL cholesterol, summary statistics will be calculated at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation). For changes from the start of Nesina treatment, summary statistics and the mean 95% confidence intervals will be calculated.

The individual laboratory values described above (mean and standard deviation) will be plotted. For the changes, the mean changes will be created using a bar graph.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.20.2-1 and Figures 5.20.2-1 to 5.20.2-10

# 6.0 Efficacy Tabulation and Analysis

#### 6.1 Changes in HbA1c

(1) Patients to be tabulated and analyzed

Efficacy Analysis Set

(2) Details of tabulation and analysis

For HbA1c (NGSP values), summary statistics will be calculated at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation). For changes, summary statistics and the mean 95% confidence intervals will be calculated and the paired t-test will be performed. Measured values of HbA1c (NGSP values) will be plotted and for the changes a bar graph will be created excluding the unknown category at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina

(3) Number of tables and figures

Table 6.1-1 and Figure 6.1-1

treatment and last evaluation).

# 6.2 Glycemic control achievement rate (HbA1c)

(1) Patients to be tabulated and analyzed

Efficacy Analysis Set

(2) Details of tabulation and analysis

The Glycemic control achievement rate for HbA1c (NGSP value) will be tabulated (< 7.0%,  $\ge 7.0\%$  / < 6.0%,  $\ge 6.0\%$ ) and a bar graph will be created (< 7.0%,  $\ge 7.0\%$  / < 6.0%,  $\ge 6.0\%$ ) at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation) (the unknown category will be excluded for the bar graph).

(3) Number of tables and figures

Table 6.2-1 and Figure 6.2-1

# 6.3 Changes in Fasting blood glucose level and Fasting insulin level

(1) Patients to be tabulated and analyzed

Efficacy Analysis Set

(2) Details of tabulation and analysis

For fasting blood glucose level and fasting insulin level, summary statistics will be calculated at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation). For changes, summary statistics and the mean 95% confidence intervals will be calculated and the paired t-test will be performed.

Measured values of fasting blood glucose level and fasting insulin level will be plotted and for

the changes a bar graph will be created excluding the unknown category at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation).

(3) Number of tables and figures

Tables 6.3-1 and 6.3-2 and Figures 6.3-1 and 6.3-2

- 6.4 Changes in HbA1c, etc. by Factor Probably Affecting Efficacy
  - (1) Patients to be tabulated and analyzed

Efficacy Analysis Set

(2) Details of tabulation and analysis

For changes in HbA1c (NGSP values), summary statistics and the mean 95% confidence intervals will be calculated and the paired t-test will be performed at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 24 months, and 36 months after Nesina treatment and last evaluation).

The Glycemic control achievement rate for HbA1c (< 7.0%,  $\ge 7.0\%$  / < 6.0%,  $\ge 6.0\%$ ) at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 24 months, and 36 months after Nesina treatment and last evaluation) will be tabulated at the following parameters:

- i Sex (Male, Female)
- ii Age ( $< 65 \text{ years}, \ge 65 \text{ years}$ )
- iii Age (< 75 years, ≥75 years)
- iv Concurrent renal disorder (No, Yes)
- v HbA1c (NGSP value) at the start of Nesina treatment (< 6.0%, 6.0% to < 7.0%, 7.0% to < 8.0%,  $\ge 8.0\%$ )
- vi Mean daily dose of Nesina (> 25 mg, 25 to > 12.5 mg, 12.5 to > 6.25 mg, or 6.25 mg)
- vii Concomitant diabetic drugs (α-glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, or insulin preparations)
- (3) Number of tables and figures

Tables 6.4-1 to 6.4-14

- 6.5 Changes in HbA1c, etc. in Patients with Special Demographics
  - (1) Patients to be tabulated and analyzed

Efficacy Analysis Set.

However, patients will be evaluated for Parameter (ii) in (2) Details of tabulation and analysis. Patients with moderate or higher renal impairment in the Efficacy Analysis Set.

(2) Details of tabulation and analysis

For changes in HbA1c (NGSP values), summary statistics and the mean 95% confidence intervals will be calculated and the paired t-test will be performed at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 24 months, and 36 months after

Nesina treatment and last evaluation).

The Glycemic control achievement rate for HbA1c ( $< 7.0\%, \ge 7.0\% / < 6.0\%, \ge 6.0\%$ ) at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 24 months, and 36 months after Nesina treatment and last evaluation) will be tabulated at the following parameters:

- i. Severity of renal impairment (Normal + Mild, Moderate + Severe)
- ii. Mean daily dose of Nesina (> 25 mg, 25 to > 12.5 mg, 12.5 to > 6.25 mg, or 6.25 mg)
- (3) Number of tables and figures

Tables 6.5-1 to 6.5-4

# Statistical Analysis Plan

# Nesina Tablets Special Drug Use Surveillance: Mild Type 2 Diabetes Mellitus

(Final Analysis)

Takeda Pharmaceutical Company Limited.



Version 1.0, Created on December 18, 2017

# Table of Contents

| 1.0 | Definition of Terms and Handling of Laboratory/Measured Data | 1 |
|---|---|---|
| 1.1 | Definitions | 1 |
| 1.2 | Important Identified Risks, Potential Risks, and Missing Information | .10 |
| 1.3 | Display digit | .11 |
| 1.4 | Level of Significance and Confidence Coefficient | .12 |
| 1.5 | Handling of Laboratory/Measured Data | .12 |
| 1.6 | Display Data Digit | .12 |
| 2.0 | Disposition of Patients (Patient Diagram) | .14 |
| 3.0 | Patient Demographics | .15 |
| 4.0 | Details of Treatment | .18 |
| 4.1 | Initial Dose of Nesina and Mean Daily Dose of Nesina, by Severity of Renal Impairment | .19 |
| 5.0 | Safety Tabulation and Analysis | .21 |
| 5.1 | Occurrence of adverse events and adverse drug reactions / infections | .21 |
| 5. | 1.1 Occurrence of adverse events | .21 |
| 5. | 1.2 Occurrence of adverse drug reactions / infections | .21 |
| 5. | 1.3 Important Identified Risks, Important Potential Risks, and Important Missing Information | .22 |
| 5.2 | Occurrence of Adverse Events and Adverse Drug Reactions / Infections in the Not Saf | ety |
| Anal | ysis Set | .23 |
| 5.2 | 2.1 Occurrence of Adverse Events | .23 |
| 5.2 | 2.2 Occurrence of adverse drug reactions / infections | .24 |
| 5.3 | Occurrence of Adverse Drug Reactions / Infections by Severity, Onset Period, and Outcome | .25 |
| 5.3 | Occurrence of Adverse Drug Reactions / Infections by Severity, Onset Period, and Outcome | 25 |
| 5.4 | Patient Demographics and Frequency of Adverse Drug Reactions / Infections by Treatment | .26 |
| 5.4 | Patients demographics and Frequency of Adverse Drug Reactions / Infections by Treatment | .26 |
| 5.5 | Occurrence of Adverse Drug Reactions / Infections by Age | .27 |
| 5.6 | Occurrence of Adverse Drug Reactions / Infections by Sex | .28 |
| 5.7 | Occurrence of Adverse Drug Reactions / Infections by Liver Disorder | .28 |
| 5.8 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Renal Disorder | .28 |
| 5.9 | Occurrence of Adverse Drug Reactions / Infections by Severity of Renal Impairment | .29 |
| 5.10 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Heart Disease | .29 |
| 5.11 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Heart Failure | .29 |
| 5.12 | Occurrence of Adverse Drug Reactions / Infections by Severity of Heart Failure | .30 |
| 5.13 | Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Stroke-rela | ted |
| Dise | ase 30 | |
| 5.14 | Occurrence of Adverse Drug Reactions / Infections by Mean Daily Dose of Nesina | .30 |
| 5.15 | Occurrence of Adverse Drug Reactions / Infections by Mean Daily Dose of Nesina in Patie | nts |
| with | Special Demographics (Patients with Moderate or Higher Renal Impairment) | .31 |
| 5.16 | Occurrence of Adverse Drug Reactions / Infections by Administration of Concomit | ant |

| Medication (Diabetic Drug) | 31 |
|---|---|
| Occurrence of Adverse Drug Reactions / Infections by Concomitant Medication (I | Diabetic Drug) |
| 31 | |
| Occurrence of Adverse Drug Reactions / Infections by Presence of Concom | itant Protease |
| nhibitors | 32 |
| Occurrence of Adverse Drug Reactions / Infections by Presence of Concomitant Re | enal Excretory |
| Orug 32 | |
| Change in Laboratory/Measured Data | 32 |
| 5.20.1 Vital Signs | 32 |
| 5.20.2 Laboratory Values | 33 |
| Efficacy Tabulation and Analysis | 34 |
| Changes in HbA1c | 34 |
| Glycemic control achievement rate (HbA1c) | 34 |
| Changes in Fasting blood glucose level and Fasting insulin level | 34 |
| Changes in HbA1c, etc. by Factor Probably Affecting Efficacy | 35 |
| Changes in HbA1c, etc. in Patients with Special Demographics | 35 |

# 1.0 Definition of Terms and Handling of Laboratory/Measured Data

# 1.1 Definitions

| Term | Definition |
|---|---|
| Nesina | Nesina tablet(s) is abbreviated as Nesina in this statistical analysis plan. |
| SOC | System Organ Class of MedDRA/J |
| | MedDRA/J version 20.1 is used for this document. |
| HLGT | High level group term of MedDRA/J |
| PT | Preferred term of MedDRA/J |
| LLT | Lowest level term of MedDRA/J |
| Registered patients | Patients whose registration was approved |
| Survey sheet (electronic) | Patients whose survey sheets were sent via GCI |
| collected patients | |
| Survey sheet (electronic) | Of the registered patients, patients whose survey sheets (electronic) were |
| uncollected patients | uncollected. |
| Safety Analysis Set | Of the survey sheet (electronic) collected patients, patients who were evaluated |
| | for safety analysis. |
| | For tabulation, the description of "total" means the Safety Analysis Set. |
| Not Safety Analysis Set | Of the survey sheet (electronic) collected patients, patients who were excluded |
| | from safety analysis |
| Efficacy Analysis Set | Of the Safety Analysis Set, patients who were evaluated for efficacy analysis |
| Not Efficacy Analysis Set | Of the Safety Analysis Set, patients who were excluded from the efficacy |
| | analysis |
| First date of Nesina | Of the start dates of the Nesina treatment period in patients, the earliest date is |
| treatment | defined as the first date of Nesina treatment. |
| Last date of Nesina | Of the last dates of the Nesina treatment period in patients, the latest date is |
| treatment | defined as the last date of Nesina treatment. If Nesina treatment is continued |
| | and the year, month, and date of the continued treatment period are specified, |
| | the year, month, and date of the continued treatment period are defined as the |
| | last date of Nesina treatment. If the data for the year, month, and date of the |
| | continued treatment period are missing, the following date is defined as the last |
| | date of Nesina treatment. |
| | (1) First date of Nesina treatment + 3 years (same month and date), if Nesina |
| | treatment is continued based on the survey sheet (electronic) after 36 |
| | months of treatment* |
| | (2) For other than the above, the first date of Nesina treatment + 1 year (same |
| | month and date), if Nesina treatment is continued based on the survey sheet |
| | (electronic) after 12 months of treatment** |

| Term | Definition |
|---|---|
| | For the continued treatment of Nesina, the following is considered as the |
| | "treatment to be continued:" |
| | • [End of Nesina tablet treatment] |
| | * If "No" for "Did you discontinue Nesina tablets by 12 to 36 months |
| | after the start of treatment?" |
| | ** If "No" for "Did you discontinue Nesina tablets by 12 months after the |
| | start of treatment?" |
| Adverse drug reactions, | Abbreviation of "adverse drug reactions / infections" |
| etc. | Of the adverse events, events for which causal relationship to Nesina was |
| | assessed as "Not related" by the Investigator. |
| | In this statistical analysis plan, "adverse drug reactions / infections" is used in |
| | the headings, while "adverse drug reactions, etc." is used in the sentences and |
| | tables. |
| Serious adverse events | Adverse events assessed as "serious" by the Investigator. |
| | Events described in the MedDRA coding list in the Takeda Medically |
| | Significant AE List will be handled as serious even if the Investigator assesses |
| | as "Not serious." |
| Serious adverse drug | Abbreviation of "serious adverse drug reactions / infections" |
| reactions | Of the "serious adverse events," the events for which causal relationship to |
| | Nesina was assessed as "Not related" by the Investigator |
| Number of patients with | Number of patients with adverse events or adverse drug reactions, etc. |
| events | |
| Number of events | Number of adverse events or adverse drug reactions, etc. |
| Percent of patients with | [For safety analysis calculation in the Safety Analysis Set] |
| events | The formula is: Number of patients with events / Number of Safety Analysis |
| | Set $\times$ 100. |
| | [For safety analysis calculation in the Not Safety Analysis Set] |
| | The formula is: Number of patients with events / Number of Not Safety |
| | Analysis Set × 100. |
| Percent of events | [For safety analysis calculation in the Safety Analysis Set] |
| | The formula is: Number of events / Number of the Safety Analysis Set $\times$ |
| | 100. |
| | [For safety calculation in the Not Safety Analysis Set] |
| | The formula is: Number of events / Number of Not Safety Analysis Set × |
| | 100. |
| Onset period | The formula is: Onset date of adverse events (or adverse drug reactions, etc.) – |
| | start date of Nesina treatment + 1. |

| Term | Definition |
|---|---|
| | For unknown onset date of adverse events (or adverse drug reactions, etc.), the |
| | onset period will be calculated as 1 day. However, if the start month and date of |
| | Nesina treatment are same as the onset month and date of adverse events (or |
| | adverse drug reactions, etc.), the onset period will be calculated as the start date |
| | of Nesina treatment. |
| Mild type 2 diabetes | Patients who have type 2 diabetes mellitus with HbA1c (NGSP value) of $\leq$ |
| mellitus | 7.4% at the start date of Nesina treatment |
| Patients with diabetic | Patients with any of the following complications: diabetic nephropathy, |
| complication | diabetic retinopathy, or diabetic neuropathy. |
| Patients with diabetic | Patients with complication of PT Code 10012660 (diabetic end stage renal |
| nephropathy | disease) or 10061835 (diabetic nephropathy). |
| Patients with diabetic | Patients with complication of PT Code 10012688 (diabetic retinal oedema) or |
| retinopathy | 10012689 (diabetic retinopathy). |
| Patients with diabetic | Patients with complication of PT Code 10012645 (diabetic autonomic |
| neuropathy | neuropathy), 10012676 (diabetic mononeuropathy), or 10012680 (diabetic |
| | neuropathy). |
| Patients with concurrent | Patients with concurrent disease of the Standardised MedDRA Query |
| hypertension | (hereinafter SMQ) Code 20000147 (hypertension (SMQ) narrow). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000026 (dyslipidaemia |
| dyslipidemia | (SMQ) narrow). |
| Patients with concurrent | Patients with concurrent disease of the PT code meeting the Takeda MedDRA |
| hyperuricemia | Query 20.1 (hereinafter, TMQ 20.1) (blood uric acid increased). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000005 (hepatic disorders |
| liver disorder | (narrow)). |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10019708 (hepatic steatosis). |
| hepatic steatosis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10019728 (hepatitis alcoholic). |
| alcoholic hepatitis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10008909 (chronic hepatitis). |
| chronic hepatitis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10019641 (hepatic cirrhosis). |
| hepatic cirrhosis | |
| Patients with concurrent | Patients with concurrent disease of the TMQ 20.1 (renal disease). |
| renal disorder | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10029164 (nephrotic |
| nephrotic syndrome | syndrome). |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10018364 (glomerulonephritis) |
| glomerulonephritis | or the PT Code 10018367 (glomerulonephritis chronic). |

| Term | Definition |
|---|---|
| Patients with concurrent | Patients with concurrent disease of the PT Code 10064848 (chronic kidney |
| chronic renal failure | disease) or the PT Code 10038435 (renal failure). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10007541 (cardiac |
| heart disease | disorders). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000004 (cardiac failure |
| cardiac failure | (SMQ) narrow). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000047 (myocardial |
| myocardial infarction | infarction (SMQ) narrow). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10007541 (cardiac disorders) |
| angina pectoris | and the PT Code 10036759 (prinzmetal angina), PT Code 10002383 (angina |
| | pectoris), PT Code 10058144 (postinfarction angina), PT Code 10002388 |
| | (angina unstable), or LLT Code 10065566 (microvascular angina). |
| Patients with concurrent | Patients with concurrent disease of cerebral infarction, cerebral haemorrhage, |
| stroke-related disease | subarachnoid haemorrhage, or transient ischaemic attack, described below. |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029205 (nervous system |
| disease cerebral infarction | disorders) and the PT Code 10006147 (brain stem infarction), PT Code |
| | 10008118 (cerebral infarction), PT Code 10008119 (cerebral infarction foetal), |
| | PT Code 10008034 (cerebellar infarction), PT Code 10019005 (haemorrhagic |
| | cerebral infarction), PT Code 10051078 (lacunar infarction), PT Code |
| | 10056237 (migrainous infarction), PT Code 10058571 (spinal cord infarction), |
| | PT Code 10060839 (embolic cerebral infarction), PT Code 10060840 |
| | (ischaemic cerebral infarction), PT Code 10064961 (thalamic infarction), PT |
| | Code 10067347 (thrombotic cerebral infarction), or PT Code 10069020 (basal |
| | ganglia infarction). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029205 (nervous system |
| cerebral hemorrhage | disorders) and the PT Code 10006145 (brain stem haemorrhage), PT Code |
| | 10008111 (cerebral haemorrhage), PT Code 10008112 (cerebral haemorrhage |
| | neonatal), PT Code 10008030 (cerebellar haemorrhage), PT Code 10018985 |
| | (haemorrhage intracranial), PT Code 10022840 (intraventricular haemorrhage), |
| | PT Code 10022841 (intraventricular haemorrhage neonatal), PT Code |
| | 10042365 (subdural haemorrhage neonatal), PT Code 10049236 (spinal |
| | epidural haemorrhage), PT Code 10048992 (spinal cord haemorrhage), PT |
| | Code 10050157 (cerebral haemorrhage foetal), PT Code 10052593 |
| | (meningorrhagia), PT Code 10058939 (thalamus haemorrhage), PT Code |
| | 10058940 (putamen haemorrhage), PT Code 10067057 (basal ganglia |
| | haemorrhage), PT Code 10067277 (cerebral microhaemorrhage), PT Code |
| | 10071205 (brain stem microhaemorrhage), PT Code 10071206 (cerebellar |
| | microhaemorrhage), PT Code 10072043 (central nervous system haemorrhage), |

| Term | Definition |
|---|---|
| | or PT Code 10073563 (Spinal subdural haemorrhage). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029205 (nervous system |
| subarachnoid hemorrhage | disorders) and the PT Code 10042316 (subarachnoid haemorrhage), PT Code |
| | 10042317 (subarachnoid haemorrhage neonatal), PT Code 10073564 (spinal |
| | subarachnoid haemorrhage), LLT Code 10072201 (Asymptomatic |
| | subarachnoid haemorrhage). |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029205 (nervous system |
| transient ischemic attack | disorders) and the PT Code 10044390 (transient ischaemic attack). |
| Patients with concurrent | Patients with concurrent disease of bronchial asthma, pollinosis, allergic |
| allergic disease | rhinitis, or allergic dermatitis, described below. |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10038738 (respiratory, |
| bronchial asthma | thoracic and mediastinal disorders) and the PT Code 10003553 (asthma), PT |
| | Code 10075084 (aspirin-exacerbated respiratory disease), PT Code 10003557 |
| | (asthma exercise induced), PT Code 10003559 (asthma late onset), PT Code |
| | 10041961 (status asthmaticus), PT Code 10001890 (alveolitis allergic), PT |
| | Code 10049585 (infantile asthma), PT Code 10070836 (occupational asthma), |
| | or PT Code 10064823 (asthmatic crisis). |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10048908 (seasonal allergy). |
| pollinosis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10039085 (rhinitis allergic). |
| allergic rhinitis | |
| Patients with concurrent | Patients with concurrent disease of the PT Code 10012434 (dermatitis allergic). |
| allergic dermatitis | |
| Patients with concurrent | Patients with concurrent disease of the SOC Code 10029104 (neoplasms |
| malignant tumor | benign, malignant and unspecified (incl cysts and polyps)). |
| Patients with concurrent | Patients with concurrent disease of the SMQ Code 20000194 (malignant |
| malignant tumor (narrow | tumour (SMQ) narrow). |
| sense) | |
| Patients with other | Patients with concurrent disease other than the above (diabetic complication, |
| concurrent disease | hypertension, dyslipidaemia, hyperuricaemia, liver disease, renal disease, heart |
| | disease, stroke-related disease, allergic disease, malignant tumor, or malignant |
| | tumor (narrow sense)). |
| Severity of renal | Severity of renal impairment in the patient demographic section |
| impairment | |

| Term | Definition |
|---|---|
| Age | If the start month and date of Nesina treatment is earlier than the birth month |
| | and date, calculate using the following formula: Start year of Nesina treatment |
| | - birth year - 1. If the birth month and date is earlier than or equal to the start |
| | month and date of Nesina treatment, calculate using the following formula: |
| | Start year of Nesina treatment – birth year. For unknown birth date, the birth |
| | date will be calculated as the 1st day of the birth month. |
| BMI | Calculate using the following formula: Weight (kg) / (0.0001 × Height (cm) × |
| | Height (cm)). Indicate to one decimal place rounded from two decimals. |
| Disease duration of type 2 | Calculate using the following formula: (start date of Nesina treatment - |
| diabetes mellitus (year) | diagnosis period of type 2 diabetes mellitus + 1) / 365.25. |
| | For unknown diagnosis month, calculate as January. |
| | Indicate to one decimal place rounded from two decimals. |
| Prior medication | Medications that patients were taking within 3 months before initiation of |
| | Nesina therapy. |
| Concomitant medication | Medications that patients were taking after the start date of Nesina treatment. |
| Start date of other diabetic | Calculate as the start date of survey sheet (electronic). |
| drug and concomitant | |
| medication (other than | |
| diabetic drug) | |
| End date of other diabetic | Calculate as the end date of survey sheet (electronic). |
| drug and concomitant | |
| medication (other than | |
| diabetic drug) | |
| Diabetic drugs | Drugs of the National Health Insurance (NHI) Drug List Code starting with |
| | 3969, 3961, 3962, 2492, 2499410, 2499411, 2499415, or 2499416. |
| α-glucosidase inhibitors | Drugs of the NHI Drug List Code starting with 3969003, 3969004, 3969009, or |
| | 3969102. |
| Thiazolidines | Drugs of the NHI Drug List Code starting with 3969005, 3969007, 3969100, |
| | 3969101, or 3969103. |
| Sulfonylureas | Drugs of the NHI Drug List Code starting with 3961 or 3969101. |
| Biguanides | Drugs of the NHI Drug List Code starting with 3962, 3969100, 3969104, or |
| | 3969105. |
| Rapid-acting insulin | Drugs of the NHI Drug List Code starting with 3969006, 3969008, 3969013, or |
| secretagogues | 3969102. |
| Insulin preparations | Drugs of the NHI Drug List Code starting with 2492. |
| DPP-4 inhibitors | Drugs of the NHI Drug List Code starting with 3969010, 3969011, 3969012, |
| | 3969014, 3969015, 3969016, 3969017, 3969024, 3969025, 3969103, 3969104, |
| | or 3969105. |

| Term | Definition |
|---|---|
| GLP-1 receptor agonists | Drugs of the NHI Drug List Code starting with 2499410, 2499411, 2499415, or |
| | 2499416. |
| SGLT2 inhibitors | Drugs of the NHI Drug List Code starting with 3969018, 3969018, 3969019, |
| | 3969020, 3969021, 3969022, or 3969023. |
| Combination of diabetic | Drugs of the NHI Drug List Code starting with 3969100, 3969101, 3969102, |
| drugs | 3969103, 3969104, or 3969105. |
| Other diabetic drugs | Other diabetic drugs not classified into the above diabetic drug categories |
| | (α-glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting |
| | insulin secretagogues, insulin preparations, DPP-4 inhibitors, GLP-1 receptor |
| | agonists, SGLT2 inhibitors, or combination of diabetic drugs). |
| Hypertension drugs | ARB Drugs of the NHI Drug List Code starting with the following 7 |
| | numbers: |
| | 2149039, 2149040, 2149041, 2149042, 2149044, 2149046, 2149048, |
| | 2149100, 2149110, 2149111, 2149112, 2149113, 2149114, 2149115, 2149116, |
| | 2149117, 2149118, 2149119, 2149120, 2149121, 2149122 |
| | Ca antagonists Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 2149019, 2149022, 2149027, 2149030, 2149034, 2149035, 2149037, 2149038, |
| | 2149043, 2149400, 2171006, 2171014, 2171019, 2171020, |
| | 2171021, 2171022, 2171405, 2190001, 2149114, 2149115, 2149116, 2149117, |
| | 2149118, 2149120, 2149121, 2149122 |
| | ACE inhibitors Drugs of the NHI Drug List Code starting with the following |
| | 4 numbers: |
| | 2144 |
| | Diuretics Drugs of the NHI Drug List Code starting with numbers 213 or the |
| | following 7 numbers: |
| | 2149003, 2149007, 2149012, 2149110, 2149111, 2149112, 2149113, 2149119, |
| | 2149122 |
| | α blockers Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 1234400, 214200210, 2149002, 2149015, 2149023, 2149026, 1152, 1149107, |
| | 1149114, 1149115, 2531001, 2149020 |
| | $\alpha\beta/\beta$ blockers Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 2149032, 2149018, 2123014, 2149009, 2123013, 2123003, 2149008, 2149016, |
| | 2442001, 2123011, 2149036, 2123016, 2149700, 2149031, 2149010, 2123001, |
| | 2123F01, 2149029, 2123008, 2149014, 2149021, 2149028, 2123015, 2123005, |
| | 2149025, 2123009, 2123403, 2149033, 2149011 |

| Term | Definition |
|---|---|
| | Complication of hypertension drugs Drugs of the NHI Drug List Code |
| | starting with the following numbers: |
| | 2149110, 2149111, 2149112, 2149113, 2149114, 2149115, 2149116, 2149117, |
| | 2149118, 2149119, 2149120, 2149121, 2149122, 2190101, 2190102, 2190103, |
| | 2190104 |
| | Other Drugs of the NHI Drug List Code starting with the following numbers: |
| | 2149047, 2142004, 2149001, 2149017, 2145 |
| Dyslipidaemia drugs | Statins Drugs of the NHI Drug List Code starting with the following numbers: |
| | 2189010, 2189011, 2189012, 2189013, 2189015, 2189016, 2189017, 2190101, |
| | 2190102, 2190103, 2190104 |
| | Fibrates Drugs of the NHI Drug List Code starting with the following numbers: |
| | 2183001, 2183002, 2183003, 2183004, 2183005, 2183006 |
| | EPA/DHA Drugs of the NHI Drug List Code starting with the following |
| | numbers: |
| | 2189019, 3399004 |
| | Other Drugs of the NHI Drug List Code starting with the following numbers: |
| | Dugs, other than the above, of the NHI Drug List Code starting with 218, |
| | 2900002, or 3133001. |
| Concomitant medication | Drugs other than the above (diabetic drugs, hypertension drugs, or |
| (other) | dyslipidaemia drugs). |
| Protease Inhibitor | Use the results of the drug name in the survey sheet (electronic) coded with the |
| | NHI Drug List (Appendix 1. List of Protease Inhibitors). |
| Renal excretory drugs | Use the results of the drug name in the survey sheet (electronic) coded with the |
| | NHI Drug List (Appendix 2. List of Renal Excretory Drugs). |
| Nesina treatment period | Actual treatment period from the start date to the end date of Nesina treatment. |
| (days) | However, the washout period is excluded from the treatment period. |
| | Calculate using the following formula: End of Nesina treatment – start date of |
| | Nesina treatment + 1 (grand total). |
| | (Consider the washout period.) |
| Mean daily dose of Nesina | Calculate using the following formula: Total of "daily dose of Nesina × Nesina |
| | treatment period at the relevant dose" / Nesina treatment period. For the |
| | calculation of Nesina treatment period, refer to the above. |
| | If the daily dose of Nesina is a number outside specification in the survey sheet |
| | (electronic) and is actual number, use the relevant number. |
| HbA1c (NGSP value) | The NGSP value only will be used in this analysis. |
| | For the HbA1c (JDS value), calculate using the following formula: |
| | NGSP value (%) = $1.02 \times JDS$ value (%) + $0.25\%$ |
| | The HbA1c (international standard value) will be handled as the NGSP value. |

| Term | Definition |
|---|---|
| Change in HbA1c | For HbA1c converted to the NGSP value, calculate using the following |
| | formula: Laboratory value at each testing time point - Laboratory value at the |
| | start of Nesina treatment. |
| Glycemic control | Divide the following two categories for the Glycemic control achievement rate: |
| achievement rate | HbA1c (NGSP converted value) [Unit %] |
| | NGSP (%): < 6.0, ≥6.0 / < 7.0,≥ 7.0 |
| non-HDL cholesterol | Calculate using the following formula: "Total cholesterol" - "HDL |
| | cholesterol." |
| Summary statistics | Number of patients, mean, standard deviation, minimum, first quartile, median, |
| | third quartile, and maximum. |

# 1.2 Important Identified Risks, Potential Risks, and Missing Information

| Term | sks, Potential Risks, and Missing Information Definition |
|---|---|
| Important identified risk | |
| Hypoglycemia | Adverse events of the following PT Codes (term) are defined as hypoglycemia. |
| | 10020994(Hypoglycaemia neonatal) |
| | 10040576(Shock hypoglycaemic) |
| | 10021000(Hypoglycaemic coma) |
| | 10020993(Hypoglycaemia) |
| | 10065981(Hypoglycaemic unconsciousness) |
| | 10021002(Hypoglycaemic encephalopathy) |
| | 10048803(Hypoglycaemic seizure) |
| | 10020997(Hypoglycaemia unawareness) |
| | 10077216(Hyperinsulinaemic hypoglycaemia) |
| | 10059035(Postprandial hypoglycaemia) |
| Acute pancreatitis | Adverse events of the SMQ Code 20000022 (acute pancreatitis (SMQ) narrow |
| | scope are defined as acute pancreatitis. |
| Hepatic impairment / | Adverse events of the SMQ Code 20000005 (hepatic disorders (SMQ) broad) |
| jaundice | are defined as hepatic impairment / jaundice. |
| Skin disorder including | Adverse events of the SMQ Code 20000020 (severe skin adverse reactions |
| oculomucocutaneous | (SMQ) narrow) are defined as skin disorder including oculomucocutaneous |
| syndrome | syndrome (Stevens-Johnson syndrome) / erythema multiforme. |
| (Stevens-Johnson | |
| syndrome) / erythema | |
| multiforme | |
| Rhabdomyolysis | Adverse events of the SMQ Code 20000002 (rhabdomyolysis/myopathy |
| | (SMQ) narrow) are defined as rhabdomyolysis. |
| Intestinal obstruction | Adverse events of the SMQ Code 20000105 (gastrointestinal obstruction |
| | (SMQ) narrow) or the HLGT Code 10018008 (gastrointestinal stenosis and |
| | obstruction) or HLT Code 10052736 (non-mechanical ileus) are defined as |
| | intestinal obstruction. |
| Interstitial pneumonia | Adverse events of the SMQ Code 20000042 (interstitial lung disease (SMQ) |
| | narrow) are defined as interstitial pneumonia. |
| Angioedema | Adverse events of the SMQ Code 20000024 (angioedema (SMQ) narrow) are |
| | defined as angioedema. |
| Important potential risk | |
| Infection | Adverse events of SOC Code 10021881(infections and infestations) are defined |
| | as infection. |
| Malignant tumor | Adverse events of the SOC Code 10029104 (neoplasms benign, malignant and |
| | unspecified (incl cysts and polyps)) are defined as malignant tumor. |

| Malignant tumor (narrow | Adverse events of the SMQ Code 20000194 (malignant tumors (SMQ) narrow) |
|---|---|
| sense) | are defined as malignant tumor (narrow sense). |
| Pemphigoid | Adverse events of the PT Code 10067776 (ocular pemphigoid) or 10034277 |
| | (pemphigoid) are defined as pemphigoid. |

| Term | Definition |
|---|---|
| Important missing | |
| information | |
| Cardiovascular system risk | Adverse events of the SMQ Code 20000047 (myocardial infarction (SMQ) |
| | broad) or SMQ Code 20000061 (central nervous system haemorrhages and |
| | cerebrovascular conditions (SMQ) broad) are defined as cardiovascular system |
| | risk. |
| | "Central nervous system haemorrhage and cerebrovascular conditions (SMQ) |
| | broad" includes the following SMQ classes. |
| | > 20000166(Conditions associated with central nervous system |
| | haemorrhages and cerebrovascular accidents (SMQ) broad) |
| | > 20000064(Cerebrovascular disorder haemorrhagic (SMQ) |
| | broad) |
| | > 20000063(Cerebrovascular disease ischaemic (SMQ) broad) |

# 1.3 Display digit

| Term | Definition |
|---|---|
| Percentage (%) | Percent of patients with adverse events or adverse drug reactions, etc. or percent |
| | of adverse events or adverse drug reactions, etc.: |
| | Indicate to two decimal places rounded from three decimals. |
| | Other than the above: |
| | Indicate to one decimal place rounded from two decimals. |
| Summary statistics | Mean, median, first quartile, and third quartile: |
| | Indicate one lower digit rounded from two lower digits than the digit of the |
| | to-be evaluated data. |
| | Standard deviation: |
| | Indicate two lower digits rounded from three lower digits of the to-be |
| | evaluated data. |
| | Minimum and maximum |
| | Indicate the same digit number as that of the to-be evaluated data (refer to |
| | Section 1.6). |
| p-value | Indicate to three decimal places rounded down from four decimals. |

| Term | Definition |
|---|---|
| | If the data is rounded down from four decimal places and less than 0.001, display |
| | as $p < 0.001$ . |

# 1.4 Level of Significance and Confidence Coefficient

Two-sided 5%, two-sided 95%.

# 1.5 Handling of Laboratory/Measured Data

- VISIT as described in the survey sheet will be used for data other than 12 months and 36 months after Nesina treatment.
- 12 months after Nesina treatment: data at 12 months after Nesina treatment will be used for the 12 months survey sheet (electronic) for patients who continued treatment.

For patients who discontinued treatment, data at 12 months after Nesina treatment will not be used for the 12 months survey sheet (electronic).

• 36 months after Nesina treatment: data at 36 months after Nesina treatment will be used for the 36 months survey sheet (electronic) for patients who continued treatment.

For patients who discontinued treatment, data at 36 months after Nesina treatment will not be used for the 36 months survey sheet (electronic).

• At the last evaluation: The last VISIT data within the evaluation period will be used.

# 1.6 Display Data Digit

Display digits are described as below.

| Term | Display digit | Unit |
|-----------------------------|---------------|-------|
| HbA1c | 0.1 | % |
| Fasting blood glucose level | 1 | mg/dL |
| Fasting insulin level | 0.1 | μU/mL |
| Fasting triglyceride | 1 | mg/dL |
| Total cholesterol | 1 | mg/dL |
| HDL-cholesterol | 1 | mg/dL |
| LDL-cholesterol | 1 | mg/dL |
| Non-HDL cholesterol | 1 | mg/dL |
| Systolic blood pressure | 1 | mmHg |
| Diastolic blood pressure | 1 | mmHg |
| Weight | 0.1 | kg |
| BMI | 0.1 | kg/m² |
| Age | 1 | Year |

| Disease duration of type 2 diabetes | 0.1 | Year |
|-------------------------------------|------|------|
| mellitus | | |
| Height | 1 | cm |
| Week of pregnancy | 1 | Week |
| Nesina treatment period | 1 | Day |
| Mean daily dose of Nesina | 0.01 | mg |

## 2.0 Disposition of Patients (Patient Diagram)

(1) Patients to be tabulated and analyzed

Registered patients

#### (2) Details of tabulation and analysis

The following will be tabulated: the number of registered patients, number of medical site at which patients is registered, number of patients whose survey sheets (electronic) are collected, number of patients whose survey sheets (electronic) are not collected, number of patients in the Safety Analysis Set, number of patients in the Not Safety Analysis Set, number of patients in the Efficacy Analysis Set, and number of patients in the Not Efficacy Analysis Set.

For the number of medical sites at which patients are registered, do not duplicate the same medical site with different departments.

For patients whose survey sheets (electronic) are not collected, tabulate the number of patients for each reason for not collected survey sheets.

For the Not Safety Analysis Set and Not Efficacy Analysis Set, the number of patients will be tabulated for each reason for exclusion to create the list.

The following is the handling of the decision whether patients who meet the following criteria should be evaluated:

| Criterion | Safety<br>evaluation | Efficacy<br>evaluation |
|---|---|---|
| Pre-agreement administration [found after administration] | × | × |
| Registration 15 days after the start of Nesina treatment [found after registration] | × | × |
| Nesina taking not confirmed [after the end of patient registration period] | × | × |
| No data for post-administration of Nesina | × | × |
| No efficacy data at two time points equivalent to the start of Nesina treatment and 3 months after Nesina treatment | 0 | × |
| Other than patients with mild type 2 diabetes mellitus | 0 | × |

o Included, × Excluded or not evaluated

#### (3) Number of tables and figures

Figure 2.0-1 and Table 2.0-1

# 3.0 Patient Demographics

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Each parameter will be classified by the categories described below to tabulate the number of patients and frequency.

| Parameter | Category |
|---|---|
| Sex | Male, Female |
| Age | Summary statistics |
| | < 65 years, ≥ 65 years |
| | < 75 years, ≥ 75 years |
| | < 20 years, 20 to 29 years, 30 to 39 years, 40 to 49 years, 50 to 59 |
| | years, 60 to 69 years, 70 to 79 years, $\geq$ 80 years |
| Disease duration of | |
| type 2 diabetes | Summary statistics |
| mellitus | |
| (year) | $<$ 2 years, 2 to $<$ 5 years, 5 to $<$ 10 years, $\ge$ 10 years, Unknown |
| Height | Summary statistics |
| Category of clinical | Outpatient, Inpatient |
| practice | Outpatient, inpatient |
| Pregnancy (only | No, Yes |
| females) | 110, 165 |
| Severity of renal | Normal, Mild, Moderate, Severe |
| impairment | Normal + Mild, Moderate + Severe |
| Concurrent disease | No, Yes |
| Diabetic complication | No, Yes |
| Details of diabetic | Diabetic nephropathy, diabetic retinopathy, diabetic neuropathy |
| complication | For the proportion, the number of patients with diabetic complication |
| (overlapped) | will be denominator. |
| Concurrent | No, Yes |
| hypertension | 110, 103 |
| Concurrent | No, Yes |
| dyslipidemia | 110, 103 |
| Concurrent | No, Yes |
| hyperuricemia | 110, 100 |
| Concurrent liver | No, Yes |
| disorder | 110, 100 |
| Details of concurrent | Hepatic steatosis, alcoholic hepatitis, chronic hepatitis, hepatic |

| Parameter | Category |
|---|---|
| liver disorder | cirrhosis, or other |
| (overlapped) | For the proportion, the number of with concurrent liver disorder will be |
| | denominator. |
| Concurrent renal disorder | No, Yes |
| Details of concurrent renal disorder (overlapped) | Nephrotic syndrome, glomerulonephritis, chronic glomerulonephritis, other For the proportion, the number of with concurrent renal disorder will be |
| (overlapped) | denominator. |
| Concurrent heart disease | No, Yes |
| Details of concurrent | Cardiac failure, myocardial infarction, angina pectoris, other |
| heart disease | For the proportion, the number of with concurrent heart disease will be |
| (overlapped) | denominator. |
| Concurrent cardiac failure | No, Yes |
| Severity classification | Classes NYHA I, NYHA II, NYHA III, and NYHA IV, Unknown |
| of cardiac failure | For the proportion, the number of with concurrent cardiac failure will |
| (NYHA classification) | be denominator. |
| Concurrent stroke-related disease | No, Yes |
| Details of concurrent<br>stroke-related disease<br>(overlapped) | Cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage, transient ischaemic attack For the proportion, the number of with concurrent stroke-related disease will be denominator. |
| Concurrent allergic disease | No, Yes |
| Concurrent malignant tumour | No, Yes |
| Concurrent malignant tumour (narrow sense) | No, Yes |
| Other concurrent disease | No, Yes |
| Past medical history | No, Yes, Unknown |
| Hypersensitivity predisposition | No, Yes, Unknown |
| Alcohol history (drinking alcoholic | Yes, No, Unknown |

| Parameter | Category |
|---|---|
| drinks almost on a | |
| daily basis) | |
| Smoking history | Never, Smoking, Smoked, Unknown |
| HbA1c(NGSP value) | Summary statistics |
| (at the start of Nesina treatment) | $< 6.0\%$ , $6.0\%$ to $< 7.0\%$ , $7.0\%$ to $< 8.0\%$ , $\ge 8.0\%$ , Unknown |
| | ≥7.4%, > 7.4%, Unknown |
| Weight | Summary statistics |
| BMI | Summary statistics |
| | $< 18.5 \text{ kg/m}^2, 18.5 \text{ to} < 25 \text{ kg/m}^2, 25 \text{ to} < 30 \text{ kg/m}^2, \ge 30 \text{ kg/m}^2,$ |
| | Unknown |
| | $< 25 \text{ kg/m}^2, \ge 25 \text{ kg/m}^2, \text{Unknown}$ |
| Dietary intervention | |
| (at the start of Nesina | Yes, No |
| treatment) | |
| Exercise intervention | |
| (at the start of Nesina | Yes, No |
| treatment) | |

Table 3.0-1

# 4.0 Details of Treatment

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Each parameter will be classified by the categories described below to tabulate the number of patients and frequency.

| Parameter | Category |
|---|---|
| Initial dose of Nesina | 25 mg, 12.5 mg, 6.25 mg, or other |
| Mean daily dose of<br>Nesina | > 25 mg, 25 to >12.5 mg, 12.5 to > 6.25 mg, or ≤6.25 mg |
| Nesina treatment period | Summary statistics |
| | 1 to 60 days, 61 to 136 days, 137 to 273 days, 274 to 455 days, ≥456 days |
| Administration of prior medication (diabetic drug) | No, Yes |
| Prior medications<br>(diabetic drugs) | α-glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, insulin preparations, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, combination of diabetic drugs, or other diabetic drugs For the proportion, the number of patients with "Yes" for administration of prior medication (diabetic drug) will be denominator. |
| Administration of prior medication (other than diabetic drug) | No, Yes |
| Administration of concomitant medication (diabetic drug) | No, Yes |
| Concomitant medications (diabetic drugs) (overlapped) | α-glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, insulin preparations, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, combination of diabetic drugs, or other diabetic drugs For the proportion, the number of patients with "Yes" for administration of concomitant medication (diabetic drug) will be denominator. |

| Parameter | Category |
|---|---|
| Administration of | |
| concomitant | No, Yes |
| medication | No, Yes |
| (hypertension drug) | |
| Concomitant medications (hypertension drugs) (overlapped) | ARB, Ca antagonists, ACE inhibitors, diuretics, $\alpha$ blockers, $\alpha\beta/\beta$ blockers, Complication of hypertension drugs, or other For the proportion, the number of patients with "Yes" for administration of concomitant medication (hypertension drug) will be denominator. |
| Administration of concomitant medication (dyslipidaemia drug) | No, Yes |
| Concomitant | Statins, fibrates, EPA/DHA, or other |
| medications | For the proportion, the number of patients with "Yes" for |
| (dyslipidaemia drugs) | administration of concomitant medication (dyslipidaemia drug) will be |
| (overlapped) | denominator. |
| Administration of concomitant medication (protease drug) | No, Yes |
| Administration of concomitant medication (combined with renal excretory drug) | No, Yes |
| Administration of concomitant medication (other) | No, Yes |

Table 4.0-1

# 4.1 Initial Dose of Nesina and Mean Daily Dose of Nesina, by Severity of Renal Impairment

(1) Patients to be tabulated and analyzed Safety Analysis Set

(2) Details of tabulation and analysis

Cross tabulation will be used for the initial dose of Nesina and the mean daily dose of Nesina, by severity of renal impairment.

Total and mild type 2 diabetes mellitus patients will be tabulated.

| return and third type 2 also even members pursuits with even and an arrangement | |
|---|---|
| Parameter | Category |
| Severity of renal impairment | Normal, Mild, Moderate, Severe |
| | Normal + Mild, Moderate + Severe |
| Initial dose of Nesina | 25 mg, 12.5 mg, 6.25 mg, or other |
| Mean daily dose of<br>Nesina | > 25 mg, 25 to >12.5 mg, 12.5 to > 6.25 mg, or ≤6.25 mg |

# (3) Number of tables and figures

Tables 4.1-1 and 4.1-2

# 5.0 Safety Tabulation and Analysis

# 5.1 Occurrence of adverse events and adverse drug reactions / infections

# 5.1.1 Occurrence of adverse events

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated for adverse events.

Total and mild type 2 diabetes mellitus patients will be tabulated.

| Parameter | Details of analysis |
|---|---|
| Number of patients with adverse events | Number of patients who experienced adverse events. |
| | Number of adverse events. Count as an event if the same adverse |
| Number of adverse | event (LLT) occur multiple times in a patient. |
| events | Count as different events for different LLTs even if they have the |
| | same PT. |
| Percent of patients with | |
| adverse events | Described in Section 1.1. |
| | Will be broadly divided into the SOCs and tabulated by PT in the |
| | SOCs. In case of the laboratory test-related events, type of adverse |
| | events will be broadly divided into the SOCs and HLGTs for |
| | tabulation by PT. |
| | For the SOCs, the number of patients with adverse events and |
| Type of advance avents | percent of patients with events will be described in the order of |
| Type of adverse events | SOCs agreed internationally. |
| | For the PTs, the number of adverse events and percent of events will |
| | be described in the ascending order of PT codes. Count as an event |
| | if the same adverse event (LLT) occur multiple times in a patient. |
| | Count as different events for different LLTs even if they have the |
| | same PT. |

# (3) Number of tables and figures

Table 5.1.1-1

# 5.1.2 Occurrence of adverse drug reactions / infections

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated for adverse drug reactions, etc. and serious adverse drug reactions, etc.

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of patients with | |
| adverse drug reactions, | Number of patients who experienced adverse drug reactions, etc. |
| etc. | |
| | Number of adverse drug reactions, etc. Count as an event if the |
| Number of adverse drug | same adverse drug reactions, etc. (LLT) occur multiple times in a |
| reactions, etc. | patient. |
| reactions, etc. | Count as different events for different LLTs even though they have |
| | the same PT. |
| Percent of patients with | |
| adverse drug reactions, | Described in Section 1.1. |
| etc. | |
| | Will be broadly divided into the SOCs and tabulated by PT in the |
| | SOCs. In case of the laboratory test-related events, type of adverse |
| | events will be broadly divided into the SOCs and HLGTs for |
| | tabulation by PT. |
| | For the SOCs, the number of patients with adverse drug reactions, |
| Type of adverse drug | etc. and percent of patients with adverse drug reactions, etc. will be |
| reactions, etc. | described in the order of SOCs agreed internationally. |
| reactions, etc. | For the PTs, the number of adverse drug reactions, etc. and percent |
| | of adverse drug reactions, etc. will be described in the ascending |
| | order of PT codes. Count as an event if the same adverse drug |
| | reactions, etc. (LLT) occur multiple times in a patient. Count as |
| | different events for different LLTs even though they have the same |
| | PT. |

Tables 5.1.2-1 and 5.1.2-2

# 5.1.3 Important Identified Risks, Important Potential Risks, and Important Missing Information

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated for important identified risks, important potential risks, and important missing information (described in Section 1.2).

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of patients with | Number of patients who experienced adverse events (or adverse |
| adverse events (or | drug reactions, etc.) with important identified risks, important |
| adverse drug reactions, | potential risks, and important missing information. |

| Parameter | Details of tabulation and analysis |
|---|---|
| etc.) | |
| Number of adverse events (or adverse drug reactions, etc.) | Number of adverse events (or adverse drug reactions, etc.) with important identified risks, important potential risks, and important missing information. Count as an event if the same adverse event (or adverse drug reaction, etc.) (LLT) occur multiple times in a patient. Count as different events for different LLTs even if they have the same PT. |
| Percent of patients with adverse events (or adverse drug reactions, etc.) | Described in Section 1.1. |
| Type of adverse events (or adverse drug reactions, etc.) | Will be broadly divided into the important identified risks, important potential risks, and important missing information and tabulated by PT in them. For the PTs, the number of adverse events (or adverse drug reactions, etc.) and percent of adverse events (or adverse drug reactions, etc.) will be described in the ascending order of PT codes. Count as an event if the same adverse event (or adverse drug reaction, etc.) (LLT) occur multiple times in a patient. Count as different events for different LLTs even though they have the same PT. |

Tables 5.1.3-1 and 5.1.3-2

5.2 Occurrence of Adverse Events and Adverse Drug Reactions / Infections in the Not Safety Analysis

Set

- 5.2.1 Occurrence of Adverse Events
  - (1) Patients to be tabulated and analyzed

Not Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated.

| Parameter | | er | Details of tabulation and analysis |
|---|---|---|---|
| Number of patients with adverse events | | ents with | Number of patients who experienced adverse events. |
| Number | of | adverse | Number of adverse events. Count as an event if the same adverse |

| Parameter | Details of tabulation and analysis |
|---|---|
| events | event (LLT) occur multiple times in a patient. |
| | Count as different events for different LLTs even if they have the |
| | same PT. |
| Percent of patients with | Described in Continue 1.1 |
| adverse events | Described in Section 1.1. |
| | Will be broadly divided into the SOCs and tabulated by PT in the |
| | SOCs. In case of the laboratory test-related events, type of adverse |
| | events will be broadly divided into the SOCs and HLGTs for |
| | tabulation by PT. |
| | For the SOCs, the number of patients with adverse events and |
| True of advance arounts | percent of patients with events will be described in the order of |
| Type of adverse events | SOCs agreed internationally. |
| | For the PTs, the number of adverse events and percent of events will |
| | be described in the ascending order of PT codes. Count as an event |
| | if the same adverse event (LLT) occur multiple times in a patient. |
| | Count as different events for different LLTs even though they have |
| | the same PT. |

Table 5.2-1

# 5.2.2 Occurrence of adverse drug reactions / infections

(1) Patients to be tabulated and analyzed

Not Safety Analysis Set

(2) Details of tabulation and analysis

The following will be tabulated.

| Parameter | Details of tabulation and analysis |
|---|---|
| Number of patients with | |
| adverse drug reactions, | Number of patients who experienced adverse drug reactions, etc. |
| etc. | |
| Number of adverse drug reactions, etc. | Number of adverse drug reactions, etc. Count as an event if the |
| | same adverse drug reactions, etc. (LLT) occur multiple times in a |
| | patient. |
| | Count as different events for different LLTs even if they have the |
| | same PT. |
| Percent of patients with | |
| adverse drug reactions, | Described in Section 1.1. |
| etc. | |

| Type of adverse drug reactions, etc. | Will be broadly divided into the SOCs and tabulated by PT in the SOCs. In case of the laboratory test-related events, type of adverse events will be broadly divided into the SOCs and HLGTs for tabulation by PT. For the SOCs, the number of patients with adverse drug reactions, etc. and percent of patients with adverse drug reactions, etc. will be described in the order of SOCs agreed internationally. For the PTs, the number of adverse drug reactions, etc. and percent of adverse drug reactions, etc. will be described in the ascending order of PT codes. Count as an event if the same adverse drug reactions, etc. (LLT) occur multiple times in a patient. Count as different events for different LLTs even though they have the same PT. |
|---|---|
|---|---|

Table 5.2-2

- 5.3 Occurrence of Adverse Drug Reactions / Infections by Severity, Onset Period, and Outcome
  - 5.3.1 Occurrence of Adverse Drug Reactions / Infections by Severity, Onset Period, and Outcome
    - (1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Each parameter will be categorized by the categories described below to tabulate the type of adverse drug reactions, etc.

Total and mild type 2 diabetes mellitus patients will be tabulated.

| Parameter | Category |
|---|---|
| Severity | Serious, Not serious |
| | 1 to 14 days, 15 to 28 days, 29 to 84 days, 85 to 168 days, 169 to |
| Onset period | 336 days, 337 to 504 days, 505 to 672 days, 673 to 840 days, 841 to |
| | 1008 days, ≥1009 days, or Unknown |
| Outcome | Resolved, Resolving, Not resolved, Resolved with sequelae, Death, |
| | or Unknown |

The method for tabulation of type adverse drug reactions, etc. is described below:

| Parameter | Details of tabulation and analysis |
|---|---|
| Type of adverse drug reactions, etc. | Will be broadly divided into the SOCs and tabulated by PT in the SOCs. In case of the laboratory test-related events, type of adverse events will be broadly divided into the SOCs and HLGTs for tabulation by PT. For the SOCs, the number of patients with adverse drug reactions, |

| Parameter | Details of tabulation and analysis |
|---|---|
| | etc. will be described in the order of SOCs agreed internationally. |
| | For the PTs, the number of adverse drug reactions, etc. will be |
| | described in the ascending order of PT codes. Count as an event if |
| | the same adverse drug reactions, etc. (LLT) occur multiple times in |
| | a patient. Count as different events for different LLTs even if they |
| | have the same PT. However, evaluate an event for the same LLT in |
| | accordance with the following order of priority: |
| | Onset period: earlier event |
| | Severity: Serious → Not serious |
| | Outcome: Death $\rightarrow$ Resolved with Sequelae $\rightarrow$ Not resolved $\rightarrow$ |
| | Resolving $\rightarrow$ Resolved $\rightarrow$ Unknown |

Tables 5.3-1 to 5.3-3

- 5.4 Patient Demographics and Frequency of Adverse Drug Reactions / Infections by Treatment
- 5.4.1 Patients demographics and Frequency of Adverse Drug Reactions / Infections by Treatment
  - (1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Each parameter will be categorized by the categories described below to tabulate the percent of patients with adverse drug reactions, etc.

The Fischer exact test will be used for parameters without rank data. The Mann-Whitney U test will be used for parameters with rank data. (The tests will be used for parameters with asterisk [\*].)

| Parameter | Category |
|-------------------------------|----------------------------------|
| Sex* | Male, Female |
| Age* | < 65 years, ≥65 years |
| | < 75 years, ≥75 years |
| Severity of renal impairment* | Normal + Mild, Moderate + Severe |
| Concurrent liver disorder* | No, Yes |
| Concurrent renal disorder* | No, Yes |
| Concurrent heart disease* | No, Yes |

| Parameter | Category |
|---|---|
| Details of concurrent | Cardiac failure, myocardial infarction, or angina pectoris |
| heart disease | |
| (overlapped) | |
| Concurrent cardiac | No, Yes |
| failure* | |
| Severity classification | Classes NYHA I, NYHA II, NYHA III, and NYHA IV |
| of cardiac failure | |
| (NYHA | |
| classification)* | |
| Concurrent | No, Yes |
| stroke-related | |
| disease* | |
| Mean daily dose of | > 25 mg, 25 to >12.5 mg, 12.5 to > 6.25 mg, or ≤6.25 mg |
| Nesina | |
| Administration of | No, Yes |
| concomitant | |
| medication (diabetic | |
| drug) | |
| Concomitant | $\alpha$ -glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, or insulin preparations |
| medications (diabetic | |
| drugs) (overlapped) | |
| Administration of | No, Yes |
| concomitant | |
| medication (protease | |
| drug)* | |
| Administration of | |
| concomitant | |
| medication (combined | No, Yes |
| with renal excretory | |
| drug)* | |

Table 5.4.1-1

# 5.5 Occurrence of Adverse Drug Reactions / Infections by Age

(1) Patients to be tabulated and analyzed Safety Analysis Set

(2) Details of tabulation and analysis

Age will be classified into < 65 years,  $\ge 65$  years and < 75 years, and  $\ge 75$  years for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Tables 5.5-1 to 5.5-2

- 5.6 Occurrence of Adverse Drug Reactions / Infections by Sex
  - (1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Sex will be classified into male or female for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.6-1

- 5.7 Occurrence of Adverse Drug Reactions / Infections by Liver Disorder
  - (1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent liver disorder will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.7-1

- 5.8 Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Renal Disorder
  - (1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent renal disorder will be classified into yes or no for tabulation of type of adverse

drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.8-1

# 5.9 Occurrence of Adverse Drug Reactions / Infections by Severity of Renal Impairment

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Severity of renal impairment will be classified into normal + mild or moderate + severe for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.9-1

# 5.10 Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Heart Disease

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent heart disease will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.10-1

# 5.11 Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Heart Failure

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent heart failure will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section

5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.11-1

- 5.12 Occurrence of Adverse Drug Reactions / Infections by Severity of Heart Failure
  - (1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Severity of heart failure will be classified into Class NYHA I, NYHA II, NYHA III, or NYHA IV for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.12-1

5.13 Occurrence of Adverse Drug Reactions / Infections by Presence of Concurrent Stroke-related

Disease

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concurrent stroke-related disease will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.13-1

- 5.14 Occurrence of Adverse Drug Reactions / Infections by Mean Daily Dose of Nesina
  - (1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

The mean daily dose of Nesina will be classified into > 25 mg, 25 to > 12.5 mg, 12.5 to > 6.25 mg, or  $\le 6.25$  mg for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section

5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.14-1

5.15 Occurrence of Adverse Drug Reactions / Infections by Mean Daily Dose of Nesina in Patients with

Special Demographics (Patients with Moderate or Higher Renal Impairment)

(1) Patients to be tabulated and analyzed

Patients with moderate or higher renal impairment in the Safety Analysis Set

(2) Details of tabulation and analysis

The mean daily dose of Nesina will be classified into > 25 mg, 25 to > 12.5 mg, 12.5 to > 6.25 mg, or  $\le 6.25$  mg for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.15-1

5.16 Occurrence of Adverse Drug Reactions / Infections by Administration of Concomitant Medication

(Diabetic Drug)

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Administration of concomitant medication (diabetic drug) will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.16-1

- 5.17 Occurrence of Adverse Drug Reactions / Infections by Concomitant Medication (Diabetic Drug)
  - (1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concomitant medications (diabetic drugs) will be classified into the following drugs:  $\alpha$ -glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin

secretagogues, or insulin preparations, for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.17-1

- 5.18 Occurrence of Adverse Drug Reactions / Infections by Presence of Concomitant Protease Inhibitors
  - (1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concomitant protease inhibitor will be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.18-1

5.19 Occurrence of Adverse Drug Reactions / Infections by Presence of Concomitant Renal Excretory

Drug

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

Concomitant renal excretory drug be classified into yes or no for tabulation of type of adverse drug reactions, etc.

The method for tabulation of adverse drug reactions, etc. is same as that described in Section 5.1.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.19-1

- 5.20 Change in Laboratory/Measured Data
  - 5.20.1 Vital Signs
    - (1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

For blood pressure (systolic/diastolic) and weight, summary statistics will be calculated at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation). For changes from the start of Nesina treatment, summary statistics and the mean 95% confidence intervals will be calculated.

Measured values (mean and standard deviation) of blood pressure (systolic/diastolic) and weight will be plotted. For the changes, the mean changes will be created using a bar graph.

Total and mild type 2 diabetes mellitus patients will be tabulated.

## (3) Number of tables and figures

Table 5.20.1-1 and Figures 5.20.1-1 to 5.20.1-6

# 5.20.2 Laboratory Values

(1) Patients to be tabulated and analyzed

Safety Analysis Set

(2) Details of tabulation and analysis

For laboratory values of fasting triglyceride, total cholesterol, HDL-cholesterol, LDL-cholesterol, and non-HDL cholesterol, summary statistics will be calculated at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation). For changes from the start of Nesina treatment, summary statistics and the mean 95% confidence intervals will be calculated.

The individual laboratory values described above (mean and standard deviation) will be plotted. For the changes, the mean changes will be created using a bar graph.

Total and mild type 2 diabetes mellitus patients will be tabulated.

(3) Number of tables and figures

Table 5.20.2-1 and Figures 5.20.2-1 to 5.20.2-10

# 6.0 Efficacy Tabulation and Analysis

#### 6.1 Changes in HbA1c

(1) Patients to be tabulated and analyzed

Efficacy Analysis Set

(2) Details of tabulation and analysis

For HbA1c (NGSP values), summary statistics will be calculated at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation). For changes, summary statistics and the mean 95% confidence intervals will be calculated and the paired t-test will be performed.

Measured values of HbA1c (NGSP values) will be plotted and for the changes a bar graph will be created excluding the unknown category at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation).

(3) Number of tables and figures

Table 6.1-1 and Figure 6.1-1

#### 6.2 Glycemic control achievement rate (HbA1c)

(1) Patients to be tabulated and analyzed

Efficacy Analysis Set

(2) Details of tabulation and analysis

The Glycemic control achievement rate for HbA1c (NGSP value) will be tabulated (< 7.0%,  $\ge 7.0\%$  / < 6.0%,  $\ge 6.0\%$ ) and a bar graph will be created (< 7.0%,  $\ge 7.0\%$  / < 6.0%,  $\ge 6.0\%$ ) at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation) (the unknown category will be excluded for the bar graph).

(3) Number of tables and figures

Table 6.2-1 and Figure 6.2-1

#### 6.3 Changes in Fasting blood glucose level and Fasting insulin level

(1) Patients to be tabulated and analyzed

Efficacy Analysis Set

(2) Details of tabulation and analysis

For fasting blood glucose level and fasting insulin level, summary statistics will be calculated at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation). For changes, summary statistics and the mean 95% confidence intervals will be calculated and the paired t-test will be performed.

Measured values of fasting blood glucose level and fasting insulin level will be plotted and for the changes a bar graph will be created excluding the unknown category at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after Nesina treatment and last evaluation).

(3) Number of tables and figures

Tables 6.3-1 and 6.3-2 and Figures 6.3-1 and 6.3-2

- 6.4 Changes in HbA1c, etc. by Factor Probably Affecting Efficacy
  - (1) Patients to be tabulated and analyzed

Efficacy Analysis Set

(2) Details of tabulation and analysis

For changes in HbA1c (NGSP values), summary statistics and the mean 95% confidence intervals will be calculated and the paired t-test will be performed at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 24 months, and 36 months after Nesina treatment and last evaluation).

The Glycemic control achievement rate for HbA1c ( $< 7.0\%, \ge 7.0\% / < 6.0\%, \ge 6.0\%$ ) at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 24 months, and 36 months after Nesina treatment and last evaluation) will be tabulated at the following parameters:

- i Sex (Male, Female)
- ii Age ( $< 65 \text{ years}, \ge 65 \text{ years}$ )
- iii Age (< 75 years,  $\ge 75$  years)
- iv Concurrent renal disorder (No, Yes)
- Which is the start of Nesina treatment (< 6.0%, 6.0% to < 7.0%, 7.0% to < 8.0%,  $\ge 8.0\%$ )
- vi Mean daily dose of Nesina (> 25 mg, 25 to > 12.5 mg, 12.5 to > 6.25 mg, or 6.25 mg)
- vii Concomitant diabetic drugs (α-glucosidase inhibitors, thiazolidines, sulfonylureas, biguanides, rapid-acting insulin secretagogues, or insulin preparations)
- (3) Number of tables and figures

Tables 6.4-1 to 6.4-14

- 6.5 Changes in HbA1c, etc. in Patients with Special Demographics
  - (1) Patients to be tabulated and analyzed

Efficacy Analysis Set.

However, patients will be evaluated for Parameter (ii) in (2) Details of tabulation and analysis. Patients with moderate or higher renal impairment in the Efficacy Analysis Set.

(2) Details of tabulation and analysis

For changes in HbA1c (NGSP values), summary statistics and the mean 95% confidence

intervals will be calculated and the paired t-test will be performed at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 24 months, and 36 months after Nesina treatment and last evaluation).

The Glycemic control achievement rate for HbA1c ( $< 7.0\%, \ge 7.0\% / < 6.0\%, \ge 6.0\%$ ) at each testing time point (start of Nesina treatment, 3 months, 6 months, 12 months, 24 months, and 36 months after Nesina treatment and last evaluation) will be tabulated at the following parameters:

- i. Severity of renal impairment (Normal + Mild, Moderate + Severe)
- ii. Mean daily dose of Nesina (> 25 mg, 25 to > 12.5 mg, 12.5 to > 6.25 mg, or 6.25 mg)
- (3) Number of tables and figures

Tables 6.5-1 to 6.5-4